## GENERAL PROJECT DATA

**Research Line:** Health. Nutrition. Neurosciences. Physiology of Nutrition and the Central Nervous System. Sleep Physiology. Ethnography.

**Project Title:** Neuro-Nutrition as Support for Physiological Performance and Cognitive Skills in People with Trisomy 21, Autism Spectrum Disorders, and Attention Deficit Disorder.

**Discipline:** Neurosciences. Nutrition. Neurobiology. Ethnography. Psychology. Sleep Physiology.

**Specialty:** Physiology of Nutrition. Biochemistry. Food Allergies and Sensitivities. Ethnography. Sleep Physiology. Neuropsychology. Neurobiology.

Principal Investigator: Dr. Reyes Haro Valencia

Type of Research: Prospective longitudinal study

**Project Duration:** 13 months

**Keywords:** Nutrition. Feeding. Trisomy 21. Down Syndrome. Autism. Attention Deficit Disorder. Hyperactivity. Cognitive Development. Sleep Physiology. Biochemistry. Physiology. Neurotransmitters. Sleep Disorders. Social Integration. Ethnography. Neurobiology. Quality of Life. Dysbiosis. Polysomnography. Evoked Potentials. Sociology. Neuropsychology. Neurodevelopment. Disability.

#### December 2021

## **Institutional Alignment and Project Justification**

The present project arises from the collaborative efforts of DOMUS Instituto de Autismo A.C., CTDUCA Atención Integral de Personas Down I.A.P., the Instituto Mexicano de Medicina Integral de Sueño, and researchers from the Universidad Nacional Autónoma de México (UNAM). These institutions share the commitment to develop scientific research with social impact, particularly in vulnerable populations with neurodevelopmental conditions.

The initial Neuro-Nutrition project, registered with the National Council of Science and Technology (CONACYT) under the title "Neuro-Nutrition as Support for Physiological Performance and Cognitive Skills in Individuals with Trisomy 21" (Project ID: 157118), provided results that exceeded expectations. These findings paved the way to broaden the scope of investigation and extend the benefits of nutritional intervention to other groups, including individuals with Autism Spectrum Disorders and Attention Deficit Disorder, with or without Hyperactivity (ADD/ADHD).

The current study builds on that foundation, seeking not only to confirm previous findings in individuals with Trisomy 21 but also to expand scientific and clinical knowledge in populations with ASD and ADD/ADHD, thereby contributing to improved quality of life, social inclusion, and health outcomes.

#### **SYNTHESIS**

Based on an extensive literature review, multiple genetic, immunological, metabolic, physiological, and therapeutic management affinities have been documented among individuals diagnosed with Trisomy 21 (Down Syndrome), Autism Spectrum Disorders (ASD), and Attention Deficit Disorder with or without Hyperactivity (ADD/ADHD). This project aims to help regularize altered metabolic processes and improve cognitive and behavioral skills in these populations through the design of an appropriate diet and the formulation of a specialized Dietary Supplement developed specifically to address the metabolic deficiencies of individuals with these conditions.

By removing harmful elements from the body and providing the appropriate nutrients, it is expected that participants' quality of life will improve both in their immediate social environment and in their sleep performance.

#### INTRODUCTION

According to data from the Instituto Nacional de Estadística y Geografía (INEGI) and the Secretaría de Salud (SSA), there are currently an estimated 150,000 individuals with Trisomy 21 (Down Syndrome) in Mexico. In relation to the population with Autism Spectrum Disorders (ASD), the Clínica Mexicana de Autismo estimates approximately 45,000 individuals nationwide, with an annual growth rate of 17%. Furthermore, the Programa Específico de Trastorno por Déficit de Atención (SSA Report 2001–2006) estimated 1.5 million children and adolescents with this condition, a number that could potentially double when including adults who continue to be affected.

Although individuals with Autism Spectrum Disorders (ASD) and Down Syndrome continue to be considered vulnerable minority groups in Mexico, the increasing prevalence of Attention Deficit Disorder, with or without Hyperactivity (ADD/ADHD), has made this condition an important focus of public health.

According to the 2010 National Population and Housing Census conducted by the Instituto Nacional de Estadística y Geografía (INEGI), there are 5,739,270 individuals in Mexico living with some form of physical or mental disability. Based on this data, approximately 30% of the disabled population in the country consists of individuals with Autism Spectrum Disorders, Down Syndrome, or Attention Deficit Disorder, with or without Hyperactivity (ADD/ADHD).

Despite awareness of these statistics, limited economic, scientific, and technological resources have been allocated to address the specific needs of these populations. In addition to the social vulnerability resulting from neglect, these groups share physiological and metabolic characteristics that make their clinical management highly specialized and complex.

Another common feature among these three populations is the global reliance on pharmacological treatment models, whose effectiveness is often limited unless combined with behavioral therapies. Stimulants such as methylphenidate and dextroamphetamine are among the most frequently prescribed medications for individuals with Down Syndrome, Autism Spectrum Disorders (ASD), and/or Attention Deficit Disorder with or without Hyperactivity (ADD/ADHD) (Rappley, 2005; Frohlich, Lanphear, & Epstein, 2007; Findling, 2008). These medications act directly on neurotransmitters such as norepinephrine and dopamine, which are closely associated with cognition, anxiety regulation, and satiety.

Some of the reported benefits of these medications include reduced impulsivity and hyperactivity, as well as improved concentration. However, their use has also been associated with adverse effects such as risk of dependency, fluctuations in body weight,

severe appetite disturbances (including anorexia or obesity), impaired growth, gastrointestinal problems, headaches, significant sleep disorders, marked variations in blood pressure (Rappley, 2005; Frohlich, Lanphear, & Epstein, 2007; Findling, 2008; Najib, 2008), and substantial hormonal imbalances.

The potential side effects of these medications often lead patients and their legal guardians (parents or caregivers) to discontinue their use, turning instead to multidisciplinary behavioral therapies. The limited understanding of the full scope of Trisomy 21, Autism Spectrum Disorders (ASD), and Attention Deficit Disorders (ADD/ADHD)—combined with the challenges of neurostimulant treatments and the modest effectiveness of psychological and behavioral interventions—has prompted both researchers and families to explore alternative therapeutic approaches. Increasingly, the scientific community is recognizing nutritional factors as decisive and fundamental in the development and clinical expression of these conditions (Sinn, 2008; Schnoll, 2003).

It is also important to acknowledge that society has prompted a redefinition of disability. Considering disability solely as a personal or individual attribute, detached from its broader social context, has significant implications for international taxonomies and for the standards used to evaluate functional impairments (Ferreira, 2006). For instance, the World Health Organization's International Classification of Impairments, Disabilities, and Handicaps (ICIDH) conceptualizes disability primarily as the consequence of a medical condition—essentially, a "natural" accident.

Research on different forms of disability has demonstrated that the family plays a central role in fostering behavioral and cognitive changes in affected individuals (Ramírez, 2011). Such changes may result from a variety of interventions, ranging from psychological programs to clinical protocols. However, there is a notable lack of quantitative studies specifically evaluating improvements in family quality of life derived from nutritional interventions.

The underlying issue is that, with the growing prevalence of neurodevelopmental disorders, it has become increasingly important to understand and anticipate their progression, as they affect individuals throughout the lifespan. Evidence from studies on these populations—and the challenges they face during the transition to adulthood, when many will outlive their parents and legal guardians—must inform discussions on service provision and public policy planning to ensure a better quality of life.

## **BACKGROUND - Feasibility of the Proposal**

#### **Research Extension**

The need to implement this protocol arises from the above-expected results of a 2011 research project supported by the Consejo Nacional de Ciencia y Tecnología (CONACYT) under the PROINOVA program (Project No. 157118), titled "Neuro-Nutrition as Support for Physiological Performance and Cognitive Skills in Individuals with Trisomy 21." The theoretical basis of that project was grounded in the physiological similarities observed between individuals with Autism Spectrum Disorders (ASD) and those with Trisomy 21 (Down Syndrome).

Key findings from the previous study that support extending the nutritional intervention to populations with Autism Spectrum Disorders (ASD) and Attention Deficit Disorder (ADD) included: strengthened immune function with fewer parasitic infections; improved absorption of proteins, calcium, phosphorus, and iron, resulting in higher growth rates compared to controls; healthier cholesterol and triglyceride profiles, thereby reducing cardiovascular risk; more efficient digestion and decreased chronic intestinal inflammation; and improved intestinal motility. In addition, participants demonstrated greater concentration, enhanced attention, and more socially adaptive behaviors.

Building on this evidence, and considering that the theoretical framework of the prior project already encompassed individuals with ASD, the present study aims to explicitly include them as a primary target population, alongside individuals with ADD.

## Etiology

The precise causes of Autism Spectrum Disorders (ASD), Down Syndrome, and Attention Deficit Disorder (ADD) remain unclear. Current therapeutic approaches are primarily aimed at alleviating symptoms that compromise quality of life, cognitive performance, and social integration. Although their etiology has not been fully established, these conditions are widely recognized as neurodevelopmental disorders that share significant genetic, immunological, metabolic, and gastrointestinal characteristics.

#### **Genetics**

Post-mortem brain studies examining genes associated with these disorders have highlighted immunological convergence rather than differences limited to neurodevelopmental genes. Consistently observed findings include immune system depression and elevated oxidative stress, both of which influence the type and severity of the disorder, as well as the degree of intellectual disability (Lintas, Sacco, & Perisco, 2010).

Mineral deficiencies—particularly calcium, magnesium, zinc, iron, and selenium—have also been linked to immune dysfunction.

Another critical factor involves neuronal development and microglial function. Excessive glutamate release and the presence of pro-inflammatory cytokines have been documented in post-mortem brains of individuals with Down Syndrome and ASD, leading to impaired inter-neuronal communication and disruption of long-range cortical-subcortical connections. These disruptions are strongly associated with deficits in cognition, social interaction, and sensory integration (Rubenstein & Merzenich, 2003; Courchesne & Pierce, 2005; Geschwind & Levitt, 2007; Belmonte, 2010).

#### Metabolism

Immune suppression in individuals with Down Syndrome, Autism Spectrum Disorders (ASD), and Attention Deficit Disorder (ADD) predisposes them to recurrent infections of the gastrointestinal tract, respiratory system, and ears. The use of antibiotics further disrupts the gut microbiota, exacerbating dysbiosis. This imbalance promotes Candida overgrowth, which contributes to the secretion of immunotoxins, intestinal wall damage, and inhibition of immunoglobulin A (IgA), ultimately leading to increased intestinal permeability (*leaky gut*). In Down Syndrome, intestinal sluggishness caused by hypotonia further prolongs exposure to pathogens.

These intestinal alterations impair secretin production, reducing pancreatic and hepatic enzyme release, and thereby hindering nutrient digestion and absorption. The processing of complex proteins such as casein (milk) and gluten (wheat, barley, rye, oats) is disproportionately affected, leaving peptides only partially digested. These altered peptides can cross compromised intestinal and blood–brain barriers, accumulate in the temporal lobes—critical for language and cognition—and exert opioid-like activity. Such effects contribute to mood instability, sensory alterations, sleep disturbances, respiratory depression, reduced attention, antisocial behaviors, and academic underperformance (Shaw, 2008).

Candida also interferes with carbohydrate metabolism by fermenting sugars, leading to three major outcomes:

- 1. Reduced ATP production from glycolysis/Krebs cycle, depriving specialized cells (e.g., hepatocytes, neurons, pancreatic beta cells) of energy.
- 2. Production of pentosidines, accelerating oxidative stress and impairing tissue regeneration.

3. Creation of alcoholic byproducts in the intestine, further damaging mucosa, impairing enzymatic activity, and reducing vitamin B synthesis.

## **Oxidative Stress and Allergies**

The fermentative activity of Candida in protein and carbohydrate metabolism, together with oxidative stress, has been associated with degenerative and autoimmune diseases such as Alzheimer's disease, diabetes, fibromyalgia, and multiple sclerosis. Nutritional control and targeted supplementation may significantly reduce these risks in populations with Down Syndrome, Autism Spectrum Disorders (ASD), and Attention Deficit Disorder (ADD).

The functional sensitivity of these groups also predisposes them to allergic or food sensitivity reactions, which may manifest as behavioral, psychological, and cognitive disturbances.

## **Quality of Life**

Scientific research on quality of life (QoL) has expanded considerably worldwide, ranging from Anglo-European contexts (Roy Brown, 2000) to Latin American settings (Verduzco, 2010). Disability is often conceptualized as the functional and social manifestation of an impairment, medically attributed to a natural accident or condition. However, this framework tends to overlook the subjective and socially constructed dimensions of disability (Ferreira, 2006).

Recognizing QoL within disability contexts now requires greater emphasis on social action and inclusion. Understanding the interrelationship between disability and QoL is fundamental to promoting equitable participation and overall well-being.

#### Sleep Physiology

#### **ASD and Sleep Disorders**

Studies have shown that children with Autism Spectrum Disorders (ASD) frequently experience sleep—wake disturbances, particularly irregular circadian rhythms (Gail, 2004). While many findings are derived from parent-reported questionnaires, objective assessments such as actigraphy and polysomnography have confirmed abnormalities in sleep architecture (Allik & Malow, 2006; Goldman & Souders, 2009). Reported prevalence rates of sleep disorders in ASD range from 44% to 83% (Gail, 2004).

Genetic anomalies affecting melatonin synthesis and signaling are considered central to these disturbances. Clinical studies indicate that melatonin administration can improve total sleep time, reduce sleep latency and nighttime awakenings, and enhance daytime behavior, with minimal adverse effects (Richdale, 1995; Wright, 2010; Rossignol, 2011; Leu, 2010).

#### **ADD and Sleep Disorders**

In children with suspected Attention Deficit Disorder (ADD), evaluation of sleep is crucial, as sleep disturbances can exacerbate ADD symptoms. Some children initially diagnosed with ADD may in fact present with primary sleep disorders such as sleep apnea or restless legs syndrome (Mindell, 2003). Sleep and attention are bidirectionally linked, sharing common prefrontal cortex mechanisms (Dahl, 1996; Kirov, 2004). The prevalence of sleep disturbances in ADD is higher than in both healthy controls and psychiatric controls (Ball, 1997; Stein & Corkum, 1999).

Experimental studies on sleep deprivation have confirmed that reduced sleep worsens attention and executive performance (Kim, 2011; Prihodova, 2010; Touchette, 2009). Adequate sleep, by contrast, has been associated with better motor skills, reaction times, and REM/N3 sleep architecture (Prehn-Kristensen, 2011). Meta-analyses estimate that up to 70% of children with ADD experience sleep disorders, with consequences for cognitive functioning, school attendance, parental mental health, and family dynamics (Sciberras, 2010; O'Callaghan, Meltzer, & Chiang, 2010).

Behavioral sleep interventions—such as sleep hygiene programs—have shown positive outcomes. When insufficient, melatonin supplementation may be considered, with evidence supporting the effectiveness of combining behavioral and pharmacological approaches (Weiskop, 2005; Hannah & Malow, 2009).

#### **Previous Dietary Supplements**

Historical attempts at dietary supplementation for Down Syndrome include:

- **1940s (USA, Dr. Henry Turkel):** A mix of 48 vitamins, minerals, and hormones. No proven long-term benefits were reported (Turkel, 1975).
- **1960s (Germany, Dr. Habound):** A vitamin–hormone–enzyme mix with no confirmed effectiveness (Habound, 1955).
- 1980s (USA, Dr. Ruth Harrell): A supplement of vitamins, minerals, and thyroid hormone showed preliminary IQ improvements in three Down Syndrome patients

- (Harrell, 1981), but results were not replicated. Commercial versions like "Haps Caps" remain unsubstantiated by scientific studies.
- 1990s (USA, Dixie Lawrence Tafoya): Building on Turkel's formula, MSB Plus was
  tested on her adopted daughter with Down Syndrome. Despite anecdotal
  improvements, it lacked scientific support. The product evolved into MSB V7 (NutriChem Labs) and later NuTriVene-D (International Nutrition), now marketed with
  modifications but still lacking independent clinical evidence.

For ASD and ADD populations, examples include:

- Formula One Supplement (Singapore, Autism Recovery Center): Marketed as detoxifying and calming, but without scientific validation.
- Kirkman Laboratories (USA): Offers a broad line of supplements categorized by function (antioxidant, digestive, immune, sleep, cognition/attention, etc.). Despite popularity, no peer-reviewed studies confirm their effectiveness. The company itself notes: "These nutritional statements have not been evaluated by the Food & Drug Administration. This product is not intended to diagnose, treat, cure, or prevent any disease."

#### **JUSTIFICATION**

## T-2 investigational nutritional formulation (research use only)

The T-2 investigational nutritional formulation, developed within the framework of this research, is a functional food formulated to support the nutritional management of individuals with Trisomy 21 (Down Syndrome), Autism Spectrum Disorders (ASD), and Attention Deficit Disorder (ADD/ADHD). Because of the distinctive characteristics of their immune systems, these individuals are particularly susceptible to intestinal dysbiosis, which disrupts metabolic pathways and exacerbates the biochemical imbalances inherent to these conditions. The T-2 investigational nutritional formulation provides naturally sourced nutrients in bioavailable forms that can be metabolized by dysbiotic intestines to help restore disrupted metabolic processes.

It is important to emphasize that the T-2 investigational nutritional formulation is not a complete food. Rather, it is designed as nutritional support specifically aimed at mitigating intestinal dysbiosis in individuals with the above-mentioned neurodevelopmental disorders. It is not intended as a treatment and does not seek to reduce intellectual disabilities or correct neurological deficits. For these reasons, it cannot be considered a drug or medication.

The T-2 formulation is formulated as a synergistic system, in which its specific ingredients interact to transform into bioactive forms that can be effectively absorbed by an organism compromised by dysbiosis. Its components function as precursors to one another, ensuring bioavailability in individuals with impaired metabolic function. When taken separately, these elements would not achieve the same therapeutic effect as when combined in the precise balance provided by the T-2 formulation.

## **Qualitative Description of Ingredients**

The scientific name of this sugar is 6-O- $\alpha$ -D-glucopyranosyl-D-fructofuranose, a disaccharide that occurs naturally in honey, sugar cane, beets, and certain fruits, though only in trace amounts. For this reason, it is commercially produced from food-grade sucrose through an enzymatic rearrangement that converts its glycosidic bond from 1,2-fructosyl to 1,6-fructosyl (Lina, Jonker, & Kozianowski, 2002).

While its properties are similar to sucrose, isomaltulose presents several important differences: it has approximately 50% of sucrose's sweetness, a lower melting point, and greater stability under acidic conditions, making it more resistant to microbial fermentation. Isomaltulose is absorbed more slowly than sucrose and is completely hydrolyzed in the small intestine, resulting in lower plasma glucose and insulin peaks. A 1985 study conducted at the University of Tsukuba showed that plasma glucose following isomaltulose ingestion rose gradually over 60 minutes to 110.9 mg/dl and then remained stable for two hours. By contrast, sucrose ingestion produced a rapid peak of 143.3 mg/dl within 30 minutes, followed by a sharp decline. These results were consistent even among individuals with diabetes, supporting isomaltulose as a suitable sweetener for this population (Kawai, Okuda, & Yamashita, 1985).

The complete hydrolysis of isomaltulose in the small intestine has been further demonstrated in urinary excretion studies, confirming that its breakdown products, glucose and fructose, are fully metabolized and absorbed (Menzies, 1974).

Isomaltulose has been extensively studied, with findings demonstrating that its consumption promotes fat oxidation both at rest and during exercise, thereby sparing glycogen reserves and reducing body fat mass without compromising systemic function (König, Theis, Kozianowski & Berg, 2011).

Further studies conducted at the University of Sydney reported that Isomaltulose has a glycemic index of 32, classified as *very low*, and provides sustained energy without abrupt glucose fluctuations. Its hydrolysis in the small intestine occurs four to five times more slowly than that of sucrose, prolonging energy release.

Because of these properties, Isomaltulose is widely used in sports nutrition, diabetic-friendly foods, and as a sucrose substitute. It does not ferment in the gut, thereby avoiding bacterial overgrowth—particularly of *Candida*—and enhances nutrient absorption when consumed in solution.

## **Whey Protein Concentrate**

Proteins are essential nutrients, second only to water in abundance in the human body. They are the fundamental components of muscles, vital organs, blood cells, enzymes, and hormones (Herman, 2009). Structurally, proteins are chains of amino acids; there are 20 in total, 9 of which are essential and must be obtained from the diet.

Animal-based proteins typically provide all essential amino acids in balanced proportions, whereas plant-based proteins require careful combination to achieve adequacy. Protein quality is evaluated through indices such as Biological Value (BV) and the Protein Digestibility Corrected Amino Acid Score (PDCAAS), the latter having been the preferred method of assessment by both the FDA and WHO since 1993.

The primary role of protein is to support tissue repair and maintenance. When consumed in excess, protein can also serve as a precursor for energy production through the Krebs cycle (Meléndez-Hevia, Waddell & Cascante, 1996). Conversely, insufficient intake compromises tissue integrity.

In individuals with Down Syndrome, Autism Spectrum Disorders (ASD), or Attention Deficit Disorder (ADD), metabolic deficiencies—including allergies or sensitivities—may impair the hydrolysis of certain animal proteins (such as casein, albumin, and red meat proteins) as well as plant proteins like gluten (Shaw, 2008).

The whey protein incorporated into the T-2 investigational nutritional formulation provides all essential amino acids with high bioavailability and closely resembles the composition of human breast milk, making it highly efficient and particularly beneficial for individuals with intestinal dysbiosis. As a pure whey protein concentrate, it carries no allergenic risk.

#### Flaxseed

The use of flaxseed as a functional food dates back centuries, particularly in European bread-making traditions. Modern studies in the United States have confirmed its health benefits. Flaxseed varieties suitable for human consumption include brown and golden,

with an average composition of 41% fat, 20% protein, 28% dietary fiber, 7.7% moisture, and 3.4% ash (Morris, 2007).

Its protein profile is similar to soy but lacks sulfur double bonds that hinder digestion. Flaxseed oil is rich in polyunsaturated essential fatty acids, including alpha-linolenic acid (Omega-3), linoleic acid (Omega-6), and oleic acid (Omega-9). Omega-3 fatty acids are metabolized into EPA and DHA with the assistance of vitamins B3, B6, C, E, and A, along with minerals such as magnesium and zinc. EPA supports the production of anti-inflammatory prostaglandins, while DHA serves as a structural component of the brain, retina, and sperm, and is a precursor to neurotransmitters such as serotonin and acetylcholine. In contrast, Omega-6 metabolism leads to arachidonic acid and pro-inflammatory prostaglandins, which must be balanced by Omega-3 derivatives (Schmidt, 1997).

Western diets often present an Omega-6 to Omega-3 ratio of approximately 20:1, inadequate for optimal EPA and DHA synthesis, and potentially contributing to the prevalence of cardiovascular diseases. Beyond its fatty acids, flaxseed provides soluble and insoluble fiber, which promotes satiety, supports glucose regulation, improves bowel motility, and contributes to lipid reduction (Morris, 2007).

Flaxseed also contains phenolic compounds with antioxidant activity, including phenolic acids, flavonoids, and lignans, which have been studied for their role in cancer prevention (Jacobs & White, 1998; Sonnenberg & Müller, 1993; Kune et al., 1998). Another component, gamma-tocopherol, acts as an antioxidant, supports blood pressure regulation, and may help prevent cardiovascular disease, cancer, and Alzheimer's disease (Chandan, Savita & Sashwati, 2006; Daun & Przybylski, 2000; Morris et al., 2005).

In addition, flaxseed contains vitamins C, B-complex, carotenoids, vitamin E isoforms, and vitamin K, which is essential for blood clotting and bone mineralization (Berkner & Runge). Its mineral profile includes calcium, copper, magnesium, manganese, phosphorus, potassium, sodium, and zinc.

The flaxseed incorporated into the T-2 investigational nutritional formulation is milled golden flaxseed and is sourced from golden flaxseed harvested at peak maturity. Its specialized processing preserves fat micelles and maximizes antioxidant content, particularly lignans, providing 10 mg per gram, equivalent to approximately 30% of the daily antioxidant requirement. Milled golden flaxseed also offers a favorable Omega-6 to Omega-3 ratio (2:3), which supports neurotransmitter production and contributes to overall metabolic balance.

#### Milk Serum Mineral Complex

Calcium is a vital mineral, with 99% of the body's stores located in bones and teeth. It also plays an essential role in muscle contraction, blood clotting, and nerve transmission. Inadequate calcium intake during childhood and adolescence compromises bone development, as nearly half of total bone mass is formed during these life stages.

The calcium included in the T-2 investigational nutritional formulation is obtained through ultrafiltration of milk serum, a process that preserves its natural nutrient balance. Its composition closely resembles that of human bone. The FDA has recognized several health claims for milk-serum mineral complex, including its role in promoting bone health, supporting postmenopausal women, enhancing calcium absorption, and preventing osteoporosis (Ward, 2007).

Milk-serum mineral complex also demonstrates high solubility in acidic environments, ensuring superior bioavailability. This enhances cellular nutrient uptake and potentiates the absorption of other nutrients present in the T-2 formula.

## **Short-Chain Fructooligosaccharides (scFOS)**

Short-chain fructooligosaccharides (scFOS) are composed of fructose molecules with a terminal glucose unit. They occur naturally in foods such as onions, asparagus, garlic, oats, rye, and artichokes, and are resistant to digestion in the upper gastrointestinal tract. Once they reach the colon, they are fermented by the microbiota and act as prebiotics.

Human studies have demonstrated that scFOS intake can increase bifidobacteria populations up to tenfold, while simultaneously suppressing pathogenic microorganisms such as Clostridia and Candida (Molis et al., 1996; Mitsuoka, Hidaka & Eida, 1987). Their prebiotic role has been formally recognized by both the World Health Organization (WHO) and the Food and Agriculture Organization (FAO) (2001), highlighting their contribution to gut health through selective microbial modulation.

Additional benefits of scFOS include enhanced absorption of calcium, magnesium, and copper (Van Den Heuvel et al., 1999; Tahiri et al., 2001; Ducros et al., 2005).

The scFOS incorporated into the T-2 investigational nutritional formulation is derived from sucrose oligomers through enzymatic processes using non-GMO Aspergillus japonicus.

More than 200 studies have confirmed that scFOS promotes the growth of bifidobacteria and lactobacilli, restores intestinal balance, enhances nutrient absorption, and improves mineral utilization. It has also been shown to support cholesterol and triglyceride reduction, accelerate gastrointestinal transit, and contribute to overall health.

#### Lactoferrin

Lactoferrin is a globular glycoprotein (peptide) responsible for transporting and delivering iron to cells, thereby regulating the presence of free iron in the bloodstream and in biological secretions. It exists in two forms: holo-lactoferrin (iron-saturated) and apo-lactoferrin (iron-free) (Levay & Viljoen, 1995).

Beyond its role in iron binding and transport, lactoferrin can also associate with other metals such as copper, zinc, manganese, gallium, and vanadium (Davidson & Lönnerdal, 2007). Its affinity for iron is approximately 300 times greater than that of transferrin, another plasma glycoprotein that regulates iron levels in biological fluids. This affinity increases in acidic environments, explaining its interaction with transferrin during inflammatory processes, when tissue pH decreases due to the secretion of lactic acid and other metabolites.

Lactoferrin is a critical component of the immune system owing to its bactericidal, fungicidal, and antiviral properties. It is present on mucosal surfaces and constitutes a major component of several secretions, including bile, saliva, pancreatic fluid, and semen, making it a key element of epithelial defense barriers. Numerous studies have demonstrated its effectiveness in combating intestinal infections caused by *Escherichia coli*.

Its antimicrobial activity is linked to its ability to sequester iron, acting as a natural bacteriostatic agent. In addition, lactoferrin exerts direct microbicidal effects by damaging microbial membranes through cytoplasmosis, thereby impairing permeability and disrupting cellular respiration in pathogens.

Although its fungicidal properties are less extensively studied, lactoferrin is known to combat Candida infections by acting synergistically with leukocytes to inhibit fungal reproduction. Its antiviral activity is primarily achieved by blocking viral attachment to host cells, thereby preventing entry and replication. This effect has been documented against several viruses, including hepatitis, rotavirus, leukemia viruses, and herpes.

Humans receive their highest dose of lactoferrin through colostrum, the first maternal milk produced after childbirth. Human milk contains the greatest concentration of lactoferrin of all mammalian milks, with colostrum containing approximately three times more than mature milk (Nagasawa, Kiyosawa & Kuwahara, 1972). After human milk, cow's milk provides the next richest source.

The lactoferrin included in the T-2 investigational nutritional formulation is sourced from cow's milk. It is extracted from whey using a process that preserves its bioactivity. Documented properties include immune modulation, stimulation of intestinal cell growth,

antimicrobial action, iron transport, inhibition of intestinal dysbiosis, and suppression of fungal overgrowth in the oral and gastrointestinal tract (Ward, 2006).

## **Pyridoxine Hydrocloride (Vitamin B6)**

Vitamin B6, also known as pyridoxine, is one of the eight vitamins in the B-complex group. Collectively, B vitamins are essential for converting carbohydrates into glucose—the body's primary energy source via the Krebs cycle—and are also involved in lipid and protein metabolism.

Specifically, Vitamin B6 plays a central role in brain development and function. It serves as the primary cofactor for the enzymes delta-5-desaturase and delta-6-desaturase, which are required for the breakdown of omega-6 and omega-3 fatty acids into critical neurotransmitters, including serotonin, epinephrine, norepinephrine, dopamine, melatonin, and gamma-aminobutyric acid (GABA). Together with Vitamin B12, it is also indispensable for the production of erythrocytes (red blood cells) and leukocytes (white blood cells), the latter being key components of the immune system.

Vitamin B6 is metabolized primarily in the liver, jejunum, and ileum, exerting much of its activity through the digestive system before being distributed to other tissues. Functionally, it acts as a coenzyme in the synthesis of hemoglobin, histamine, neurotransmitters, and in the metabolism of lipids, glucose, and amino acids.

The T-2 formulation includes pyridoxine hydrochloride (vitamin B6).

## Systemic Functioning of the T-2 investigational nutritional formulation

The T-2 investigational nutritional formulation acts on multiple metabolic pathways and biochemical processes, not only through the properties of its individual components but also through their synergistic interactions, which enhance systemic balance across organs and tissues.

Isomaltulose, being enzymatically rather than bacterially hydrolyzed, is not a viable substrate for pathogenic microorganisms such as *Candida*. This property reduces parasitic colonization throughout the gastrointestinal tract and helps prevent nutrient malabsorption. In combination with lactoferrin, which provides antimicrobial protection at entry points such as the oral cavity, the investigational formulation establishes protective conditions from ingestion onward.

The strong glycosidic bond of Isomaltulose ensures sustained energy release, avoiding abrupt glucose spikes and subsequent hypoglycemic crashes. Unlike sucrose, which is rapidly fermented by bacteria, Isomaltulose supports a balanced supply of glucose and glycogen, stabilizes insulin secretion, and reduces anxiety, thereby contributing to improved learning, concentration, emotional regulation, and appetite control.

Its synergy with milled golden flaxseed flaxseed further promotes fat metabolism by encouraging the body to utilize fat reserves when carbohydrate absorption is slowed. Together, Isomaltulose, flaxseed, and scFOS promote the restoration of intestinal balance by stimulating the growth of beneficial bifidobacteria and lactobacilli, improving nutrient absorption, and optimizing osmolarity (170–295 mOsm/L).

Whey protein concentrate whey protein supports the repair of intestinal lesions caused by *Candida* and *Clostridia*. This is particularly relevant given that the small intestine produces up to 95% of the body's serotonin and 50% of its dopamine (Manocha et al., 2012; Gershon, 1999; Mirre, 2012). By restoring intestinal integrity, Whey protein concentrate enhances neurotransmitter production, with synergistic effects amplified by milk-serum mineral complex calcium and flaxseed-derived vitamin K, both of which are essential for bone health and blood coagulation.

Milled golden flaxseed flaxseed provides 1.09 g of dietary fiber per serving, which contributes to improved intestinal motility and helps maintain microbiota balance. Its fatty acid profile ensures the sequential metabolic conversion of oleic acid (omega-9), linoleic acid (omega-6), and alpha-linolenic acid (omega-3) into arachidonic acid, EPA, DHA, and prostaglandins, thereby supporting inflammatory regulation and cerebral blood flow.

#### **Dosage and Administration**

Participants will be instructed to take 23 g of the T-2 investigational nutritional formulation, twice daily, dissolved in 250 ml of liquid.

For the study population (Trisomy 21, ASD, and ADD/ADHD), it is recommended that the investigational formulation be prepared with Casein-free beverage, which is casein-free and enriched with probiotic fiber. However, it may also be consumed with other liquids—including cow's milk, plant-based beverages, coffee, tea, water, or natural juice—without altering its properties. The formulation can be taken hot, cold, or warm.

The first daily dose should be consumed upon waking, ideally 30–60 minutes before breakfast. The second dose should be taken in the afternoon, approximately two hours before sleep, regardless of dinner timing.

## **Ethnography**

Studying quality of life (QoL) in families with a member diagnosed with Autism Spectrum Disorders (ASD), Attention Deficit Disorder (ADD/ADHD), or Trisomy 21 (Down Syndrome) is a central aspect of this research. Such analysis makes it possible to assess not only the progress of participants undergoing nutritional intervention but also the broader impact on family dynamics.

In recent years, QoL has gained increasing importance due to the limited opportunities for social, family, and leisure activities, particularly in households managing neurodevelopmental conditions. Evidence from the initial phases of this line of research has demonstrated that nutritional interventions can strengthen specific abilities in individuals with disabilities while also enhancing the overall well-being of their families.

These outcomes justify expanding the scope of investigation from ethnographic exploration to sociological analysis, providing valuable insights into the cognitive and behavioral evolution of participants, as well as the adaptive changes within their families over the course of one year.

## Sleep Physiology

This study aims to evaluate a balanced dietary intervention formulated with Isomaltulose, whey protein concentrate, flaxseed, milk-serum mineral complex, scFOS, Luo Han Guo (as a natural sweetener), and lactoferrin. The impact of this intervention on children with Trisomy 21 (Down Syndrome), Autism Spectrum Disorders (ASD), and Attention Deficit Disorder (ADD/ADHD) will be objectively assessed through neurophysiological testing and blood chemistry analyses.

Given that sleep disorders are highly prevalent in these populations and that diet is known to influence symptom expression, this project also seeks to explore the interplay between diet, sleep, and behavior. By addressing this understudied area, the study aims to generate evidence that can inform more comprehensive management strategies for children with neurodevelopmental conditions.

## Neuropsychological

Down Syndrome (DS) is the most common genetic cause of intellectual disability (ID), defined as an IQ below 70. Severity is typically classified as mild (IQ 55–70), moderate (IQ 40-54), severe (IQ 25-39), or profound (IQ < 25) (Vaillend et al., 2008). Approximately 30% of moderate to severe cases of intellectual disability are associated with DS (Stoll et al., 1990; Pulsifer, 1996).

Intellectual disability in DS impacts multiple domains, including cognitive development, language acquisition, motor skills, learning, and memory (Brown et al., 1990; 2003; Raz, 1995; Pulsifer, 1996; Hodapp et al., 1999; Chapman et al., 1998; Carlesimo et al., 1997; Clark & Wilson, 2003; Nadel, 2003; Pennington et al., 2003).

Although IQ testing has traditionally been the primary diagnostic tool, current recommendations emphasize the use of comprehensive assessments that incorporate daily living skills, cognitive processes, and emotional functioning, employing tools that are both culturally and linguistically adapted (Rondal, Perera & Spiker, 2011; Edgin et al., 2010).

#### **HYPOTHESIS**

Through a biomedical protocol involving dietary intervention and nutritional reinforcement with the T-2 investigational nutritional formulation, formulated for individuals with Down Syndrome (DS), Autism Spectrum Disorders (ASD), and Attention Deficit Disorder (ADD/ADHD), it is anticipated that intestinal dysbiosis, pathogenic burden (bacteria, fungi, yeasts), and oxidative stress will be reduced. This intervention is expected to promote a balanced nutritional state and support the production of key neurotransmitters, thereby contributing to improvements in quality of life, sleep regulation, concentration, cognition, self-regulation, and social interactions. Secondary Hypothesis

Oral administration of T-2 in mice will increase dendritic spines and synapses and improve performance in motor and cognitive tasks.

#### **OBJECTIVES**

- Improve compromised metabolic processes inherent to these conditions, as reflected in indicators such as dysbiosis, infections, food sensitivities, malnutrition, thyroid function, and neurotransmitter utilization.
- Strengthen the immune system, reducing allergies, sensitivities, otic and respiratory infections, and gastrointestinal pathogens.

- Reduce oxidative stress, leading to decreased anxiety, improved sleep quality, and enhanced Krebs cycle efficiency.
- Enhance gastrointestinal function and nutrient absorption, assessed through markers such as reflux, cholesterol and triglyceride levels, bowel regularity, stool formation, and improvements in body mass index (BMI).
- Improve quality of life, including stabilization of mood, increased social interactions, and reinforcement of cognitive processes such as attention, adaptability, and concentration.

## **Secondary Objectives**

- Ethnography: Quantify the impact of the nutritional intervention on families of individuals with Trisomy 21, Autism Spectrum Disorders (ASD), and Attention Deficit Disorder (ADD/ADHD), with particular attention to changes in family dynamics across different phases of the study.
- Sleep Physiology: Investigate the relationship between diet and sleep in children with ADD and ASD, evaluating the effectiveness of dietary modification on sleep patterns and expression.

# CONTRIBUTION OF THE PROJECT TO ADVANCING KNOWLEDGE IN ITS OWN FIELD AND AREA OF RESEARCH

This project represents the first biomedical protocol in Mexico to investigate neuro-nutrition—defined as dietary intervention combined with nutritional enrichment—in populations with Autism Spectrum Disorders (ASD) and Attention Deficit Disorder (ADD/ADHD), while also expanding upon the findings previously obtained in the first stage of this protocol with individuals with Trisomy 21 (Down Syndrome).

The primary aim is to provide both quantitative and qualitative evidence that disability in individuals with DS, ASD, and ADD extends beyond intellectual impairment into biological domains.

The project further seeks to enhance understanding of the metabolic and physiological characteristics of these populations, thereby informing the design of appropriate therapeutic management strategies.

Finally, it intends to demonstrate that ADD encompasses neurobiological, electrical, and biochemical processes, extending beyond the psychosocial dimensions traditionally emphasized.

#### **METHODOLOGY**

## **Operational Duration**

The project will run for a period of 13 months.

## **Population Description**

The estimated total population is 72 individuals between 2 and 35 years of age, divided into three groups based on their neurodevelopmental condition:

- Trisomy 21 (Down Syndrome, DS)
- Autism Spectrum Disorder (ASD)
- Attention Deficit Disorder (ADD)

Each group included between 24 and 27 participants, with more males than females. Ages ranged from 2–33 years for ASD, 2–30 years for DS, and 5–14 years for ADD. Mean ages and BMI values are shown in Table 1.

| Participants | ASD<br>(N = 27) | | DS<br>(N = 24) |
|---|---|---|---|
| • | Mean (SD) | Mean (SD) | Mean (SD) |
| Age (years) | 2-33<br>11.51±8.5 | 5-14<br>8.8±2.32 | 2-30<br>13.7±7.25 |
| Body mass index (kg/m <sup>2</sup> ) | 19.11±3.71 | 18.41±4.01 | 21.92±6.27 |
| Men | 24 | 20 | 14 |
| Women | 3 | 5 | 10 |

Table 1. Characteristics of each group

For participants with Autism Spectrum Disorders (ASD), recruitment was conducted at DOMUS Instituto de Autismo A.C., where diagnoses were confirmed using DSM-IV criteria (First et al., 2002). Symptom severity was assessed with the IDEA (Inventario del Espectro Autista-Autism Spectrum Inventory), which evaluates 12 developmental dimensions across four areas and is scored on a scale from 0 to 8. Scores between 70–96 indicate classic Kanner autism, 50–70 correspond to regressive autism, 40–50 reflect high-functioning

autism, and 30–45 indicate Asperger's syndrome (Martos & Morueco, 2007; García-López & Narbona, 2014b). The mean IDEA score for this sample was 63 ± 18 (Table 2).

| Diagnostic (DSM-IV) | IDEA (Autism Spectrum Inventory) |
|---|---|
| ASD N = 27 | Classic Kanner Autism (70–96) – 40% |
| Pervasive Developmental Disorders (PDD): | "Regressive Autism" (50–70) – 40% |
| Autistic Disorder – 74% | High-Functioning Autism (40–50) – 4% |
| Pervasive Developmental Disorders, Not | A a m a w g a w a d w a m a (20, 45), 100/ |
| Otherwise Specified (PDD-NOS) – 26% | Asperger's Syndrome (30–45) – 16% |

Table 2. Diagnosis and IDEA scores in ASD participants

For participants with Attention Deficit Disorder (ADD/ADHD), recruitment was conducted through schools specializing in this condition. Diagnosis was confirmed using the Conners' Parent Rating Scale – Revised (Long Form), which assesses behavioral and learning difficulties, psychosomatic complaints, impulsivity, hyperactivity, and anxiety (Conners, 1999). The Hyperactivity Index was applied, with scores greater than 16 for boys and 12 for girls aged 6–11 indicating clinically significant hyperactivity (Orjales Villar, 1998) (Table 3).

| Check list DSM-IV | Hyperactivity Index | |
|-------------------|----------------------------|------|
| | Conners Revised Scale | |
| ADD | Girls (n=4) with suspected | 50 % |
| N = 25 | ADD (>12) | |
| | Boys (n=21) with suspected | 33 % |
| | ADD (>16) | |

Table 3. Conners' Scale results for ADD participants

For DS, participants came from "CTDUCA Atención Integral de Personas Down IAP" and "Integración Down IAP." All had karyotype-confirmed diagnoses, with one case of mosaicism.

## **Population Segregation**

Each diagnostic group was further divided into three subgroups:

- Pilot Group: Received 23 g of T-2 twice daily and followed a strict dietary intervention protocol.
- Diet Group: Followed the dietary intervention protocol without supplementation.
- Control Group: Received neither supplementation nor dietary intervention.

The study population (ages 2–35) was further stratified into subgroups A–G (3–30 years) according to developmental stages (*Figure 6: Age distribution*).

| Subgroup | Lower limit | Upper limit |
|----------|-------------|-------------|
| А | 3 | 5 |
| В | 6 | 9 |
| С | 10 | 13 |
| D | 14 | 17 |
| Е | 18 | 21 |
| F | 22 | 25 |
| G | 26 | 30 |

Figure 6. Population distribution by age groups

#### **Clinical Evaluation**

Clinical follow-ups included parental reports and physical examinations aimed at detecting allergies, food sensitivities, candidiasis, infections, gastrointestinal disturbances, chronic otitis media, and other recurrent conditions. A 25-item checklist was applied, covering digestive, respiratory, dermatological, and systemic indicators.

## **Laboratory Studies**

Laboratory support included:

- Blood count: red/white series, platelets, sedimentation.
- Blood chemistry: glucose, urea, creatinine, uric acid, lipids, triglycerides.
- C-reactive protein: marker of inflammation.
- Serum homocysteine: marker of fat metabolism and oxidative stress.
- Plasma cortisol: indicator of adrenal activity.
- Thyroid panel: T4, free T4, T3, protein-bound iodine, TSH, total cholesterol.

• Stool analyses: coprological, coproparasitoscopic (3 samples).

Some specialized biochemical analyses were conducted at The Great Plains Laboratory (Kansas, USA), led by Dr. William Shaw, including:

- IgG Food Allergy Panel (93 foods).
- Comprehensive Organic Acid Test (65 metabolites).
- Urinary peptides from gluten and casein.

## **Anthropometrics**

Weight, height, and BMI were measured monthly, compared against WHO growth standards (BMI-for-age) and Mexican NOM references (NOM-008-SSA2-1993; NOM-174-SSA1-1998).

## **Ethnography**

The study adopted a longitudinal approach using the Sherlock model, combining quantitative and qualitative assessments of personal, functional, and social quality of life. Families underwent three structured interviews (baseline, mid-study, final), recorded in audio and video, with statistical and content analysis applied to results.

#### Neuropsychology

**IDEA Inventory (ASD):** Applied to establish severity, guide interventions, and assess treatment impact across 12 dimensions.

**Down Syndrome:** Cognitive assessments emphasized daily life skills, cognitive processes, and emotional capacities. Recommended tests were culturally and linguistically adapted (Rondal, Perera & Spiker, 2011; Edgin et al., 2010). Tools included:

- Ages 3–6: BATELLE developmental inventory (Newborg et al., 1998).
- Ages 6–35: NEUROPSI Attention and Memory (Ostrosky et al., 2003), Executive Function Battery (Flores et al., 2008, 2011), computerized neuropsychological tasks (Ostrosky et al., 2003), basic emotion recognition tasks, Barthel Index (Cid-Ruzafa & Damián-Moreno, 1997), and BRIEF executive function scale (Goia et al., 2000).

The neuropsychological evaluation was coordinated by Dr. Maura Jazmín Ramírez Flores, with support from trained psychology interns (4–6 students).

**ADD:** NEUROPSI Attention and Memory (6–85 years), EDAH (for ADHD), and Conners' Scales (long parent version, 80 items) were applied.

#### Polysomnography and P300

Polysomnographic assessments included recordings of EEG, EOG, EMG, heart rate, respiratory effort, airflow, oxygen saturation, limb movements, and sleep architecture. Data were analyzed according to international standards and compared with control groups using ANOVA.

Measured variables included total sleep time, wake time, sleep efficiency index, distribution of sleep stages, number of awakenings, apnea-hypopnea index, and periodic limb movement index. Additionally, P300 event-related potentials were incorporated as an independent clinical measure.

All studies were conducted at a specialized sleep clinic in Mexico City, and participants received dietary support throughout the study period.

## **Family Seminars**

To support families and disseminate the objectives of the study, a series of educational seminars was organized. Topics addressed included candidiasis, allergies, biomedical protocols, psychological adaptation to disability, family dynamics, and nutritional interventions (e.g., gluten-free diets, food additives, and cooking classes).

The sessions were delivered by Dr. Javier Hernández Covarrubias, Psychologist María Angélica Núñez, and Biochemical Engineer Cecilia Fernández Aguirre.

#### BENEFITS AND RISKS FOR THE POPULATION

This is considered a minimal-risk study, as supplementation does not pose a health risk and does not involve pharmaceutical compounds.

Risks associated with sample collection, electrophysiological studies, and psychological testing will be managed by the professional staff of the Instituto Mexicano de Medicina Integral de Sueño. In all cases, follow-up will be provided by a multidisciplinary medical

team that includes specialists in Otorhinolaryngology, Psychology, Geriatrics, Dentistry, Pediatrics, Neurology, Psychiatry, Pulmonology, and Internal Medicine.

All participants will receive reports from their clinical assessments, evaluations, and electrophysiological studies, along with specialized counseling. Any conditions requiring medical care will be addressed and followed up by qualified medical professionals.

#### ASSIGNMENT OF RESPONSIBILITIES: RESEARCH TEAM AND ASSOCIATED ENTITIES

#### **Professional Staff**

- Dr. Reyes Haro Valencia Principal Investigator (CONACYT CVU: 74747)
- Dr. Elizabeth Ibarra Coronado Sleep Physiology Area Leader (CONACYT CVU: 288056)
- I.Q.I. Edilberto Sánchez Technical Coordinator (CONACYT CVU: 392429)
- Eng. Miguel Hidalgo Olvera Legal Representative and Administrative Coordinator (CONACYT CVU: 392684)
- Lic. Mónica Matilde Apodaca Aragón Project Administrator (CONACYT CVU: 499625)
- I.B. Cecilia Fernández Aguirre Biomedical Area Leader (CONACYT CVU: 353604)
- Dr. Octavio César García González Neurobiology Area Leader (CONACYT CVU: 39694)
- Dr. Maura Jazmín Ramírez Flores Neuropsychological Evaluation for Down Syndrome (CONACYT CVU: 174346)
- Lic. Juana Elvira Portillo Navarro Neuropsychological Evaluation for ADD (CONACYT CVU: 510484)
- Arturo Ramírez Ramos Ethnographic Area Leader (CONACYT CVU: 510634)

#### Institutional Site

Instituto Mexicano de Medicina Integral de Sueño

#### **Associated Entities**

- Mexico: Olarte y Akle Bacteriólogos, S.A. de C.V.
- United States: The Great Plains Laboratory, Inc.

Integración Down, I.A.P.

• Domus Instituto de Autismo

#### **PROGRESS CONTROL PLAN**

The project is scheduled to last 13 months, from December 2021 to December 2022, and will be divided into two stages of approximately six months each.

## Stage I: Design and Intellectual Property Protection

**Duration:** First Semester

## **Objectives:**

• Confirm the physiological and metabolic similarities documented in the literature across the study populations and design a unified nutritional intervention scheme.

• Determine expected cerebral modifications resulting from the intervention by standardizing the protocol in neurotypical animal models.

#### Goals:

 Create a homogeneous information base documenting physiological and metabolic affinities among the target populations.

• Obtain audiovisual records of families highlighting quality of life aspects.

• Establish a specialized dataset on sleep habits of individuals with the studied neurodevelopmental disorders.

 Document neuropsychological and behavioral profiles within family, social, and school contexts.

#### **Activities:**

• Bimonthly 1: Confirm study populations (Down Syndrome, ASD, ADD).

Assign dietary subgroups (Pilot, Diet, Control).

• Conduct studies of the T-2 investigational nutritional formulation

 Baseline studies including laboratory tests, clinical reviews, anthropometric measures, ethnographic interviews, neuropsychological tests, full polysomnographic records, and P300 potentials. • Standardize animal model protocol.

• **Month 1:** Start nutritional intervention (diet implementation).

 Month 4-6: Report baseline results, documenting biomedical, dietary, familial, cognitive, behavioral, and sleep-related findings. Conduct behavioral tests in animal

models.

**Expected Results at the End of Stage I (6 months):** 

Statistical report on physiological profiles, allergies, and food sensitivities.

Statistical report on sleep disorders and comorbidities.

Repository of family testimonies on quality of life.

**Stage II: Scientific Conclusions** 

**Duration:** Second Semester

Document and analyze biomedical, neuropsychological, sleep-physiology, and

ethnographic outcomes across groups.

Goals:

Validate or reject the hypothesis of cognitive and behavioral improvements following

dietary intervention, contrasting supplemented versus non-supplemented groups.

• Evaluate secondary hypotheses regarding ethnography and sleep physiology.

**Activities:** 

• Conduct follow-up studies (laboratory tests, clinical reviews, anthropometric

measures, ethnographic interviews, neuropsychological tests, polysomnography,

P300 potentials).

Report comparative analyses between baseline and follow-up results.

• Document biochemical, immunological, familial, social, and neuropsychological

changes, as well as sleep physiology outcomes.

**Expected Results and Deliverables at the End of Stage II:** 

Technical reports on biochemical, anthropometric, and dietary allergy/sensitivity

changes.

- Technical reports on changes in quality of life within families and social circles.
- Technical reports on sleep habit modifications.
- Technical reports on cognitive and behavioral changes.

#### REFERENCES

Accardo JA, Marcus CL, Leonard MB, Shults J, Meltzer LJ, Elia J. (2012) Associations Between Psychiatric Comorbidities and Sleep Disturbances in Children with Attention-Deficit /Hyperactivity Disorder. J Dev Behav Pediatr. 33(2):97-105.

Achenbach TM, Rescorla LA. (1999) Manual for the ASEBA school-age forms & profiles: an integrated system of multi-informant assessment. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families; 2001. Hering E, Epstein R, Elroy S, Iancu DR, Zelnik N. Sleep patterns in autistic children. J Autism Dev Disord. Apr;29(2):143-7.

Adesman AR, Altshuler LA, Lipkin PH, Walco GA. (1990). Otitis media in children with learning disabilities and in children with attention deficit disorder with hyperactivity. Pediatrics. 85:442-6.

Ali NJ, Pitson D, Stradling JR. (1996). Sleep disordered breathing: effects of adenotonsillectomy on behaviour and psychological functioning. Eur J Paediatr. 155:56-62.

Allik H, Larsson JO, Smedje H. (2006). Sleep patterns of school-age children with Asperger syndrome or high-functioning autism. J Autism Dev Disord. 2006;36(5):585-95.

Altman J, Das GD, Sudarshan K. 1970. Dev Psychobiol. 3 (4):281-301. The influence of nutrition on neural and behavioral development. I. Critical review of some data on the growth of the body and the brain following dietary deprivation during gestation and lactation.

Alvarez VA, Sabatini BL. 2007. Anatomical and physiological plasticity of dendritic spine. Ann. Rev. Neurosci. 30: 79-87.

American Academy of Pediatrics, Committee on Quality Improvement and Subcommittee on ADHD. Clinical practice guideline: diagnosis and evaluation of the child with attention-deficit/hyperactivity disorder. Pediatrics. 2000;105:1158-70.

American Academy of Pediatrics, Committee on Quality Improvement and Subcommittee on ADHD. Clinical practice guideline: Treatment of the school-aged child with attention-deficit/hiperactivity disorder. Pediatrics. 2001;108:1033-44. 71.

American Academy of Sleep Medicine. International Classification of Sleep Disorders, 2nd ed. Diagnostic and Coding Manual. Westchester, Illinois. American Academy of Sleep Medicine, 2005.

American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders. 4th ed. American Psychiatric Press; Washington, DC: 2000a. Text Revision

American Psychiatric Association. Diagnostic and statistical manual for mental disorders. 4th ed. DSM-IV. Washington DC: APA; 1994.

American Type Culture Collection. "Mission". http://www.atcc.org/About/tabid/138/Default.aspx

Anacleto TS, Louzada FM, Pereira EF. Ciclo vigília/sono e o transtorno de déficit de atenção/hiperatividade. Rev Paul Pediatr. 2011;29(3): 437-42.

Andrade JP, Castanheira-Vale AJ, Paz-Dias PG, Madeira MD, Paula-Barbosa MM. 1996. The dendritic tres of neurons from hippocampal formation of protein-deprived adults rats. A quantitative Golgy study. Exp. Brain Res. 109(3):419-433.

Andrade JP, Lukoyanov NV, Paula-Barbosa MM. 2002. Chronic food restriction is associated with subtle dendritic alterations in granule cells of the rat hippocampal formation. Hippocampus 12: 149-164.

Antonarakis SE, Lyle R, Dermitzakis ET, Reymond A, Deutsch S. 2004. Chromosome 21 and Down syndrome: from genomics to pathophysiology. Nat. Rev. Gent. 5: 725-738.

Arnold LE, DiSilvestro RA. Zinc in attention-deficit/ hyperactivity disorder. J Child Adolesc Psychopharmacol. 2005;15:619–627.

Arnold LE. Methylphenidate versus amphetamine: a comparative review. En: Greenhill LL, Oshman BB, editors. Ritalin: theory and practice. 2nd ed. Larchmont: Mary Ann Liebert, Inc.; 2000. p. 127-40.

Ashkenasi A. Effect of Transdermal Methylphenidate Wear Times on Sleep in Children with Attention Deficit Hyperactivity Disorder. Pediatric Neurology 2011;45(6),381-386.

Autism Recovery Centre. Multi-Vitamins & Minerals: "Formula One". Disponible en: http://autismrecovery.com.sg/formula-one-p-

84.html?zenid=d94a67e08cc4cd5107b16dfc381eda71

Avior G, Fishman G, Leor A, Sivan Y, Kaysar N, Derowe A. The effect of tonsillectomy and adenoidectomy on inattention and impulsivity as measured by the Test of Variables of

Attention (TOVA) in children with obstructive sleep apnea syndrome. Otolaryngol Hed Nek Surg. 2004;131:367-71.

Balboa, María A & Balsinde, Jesús. (2006). "Oxidative Stress and Arachidonic Acid Mobilization". Instituto de Biología Molecular y Genética. Consejo Español de Investigación y Facultad de Medicina de la Universidad de Valladolid. Biochimica et Biophysica Acta (BBA). Molecular Cell Biology of Lipids. Volume 1761, Issue 4, 385-391.

Ball JD, Tiernan M, Janusz J, Furr A. Sleep patterns among children with attention-deficit/hyperactivity disorder: a reexamination of parent perceptions. J Pediatr Psychol. 1997;22:389-98.

Barkley RA. Behavioral inhibition, sustained attention, and executive functions: constructing a unifying theory of ADHD. Psychol Bull. 1997;121:65-94.

Baron-Cohen, S. & Bolton, P., Autismo una guía para padres. Madrid, Alianza Editorial, 1998

Baron-Cohen, S.; Hadwin, J.; Howlin, P. & Hill, K., ¿Podemos enseñar a comprender emociones, creencias o ficciones a los niños autistas?. En: El Tratamiento del Autismo. Nuevas Perspectivas. Riviere & Mattos, Comp. Madrid, IMSERSO, 2001

Bartlett WP, Banker GA. 1984. An electron microscopic study of the development of axons and dendrites by hippocampal neurons in culture. Cells which develop without intracellular contacts. J. Neurosci. 4: 1944-1953.

Belichenko PV, Kleschevnikov AM, Salehi A, Epstein CJ, Mobley WC. 2007. Synaptic and cognitive abnormalities in mouse models of Down syndrome: exploring genotype-phenotype relationships. J. Comp. Neurol. 504: 329 345.

Belichenko PV, Masliah E, Kleschevnikov AM, Villar A, Epstein CJ, Salehi A, Mobley WC. 2004. Synaptic structural abnormalities in the Ts65Dn mouse model of Down syndrome. J. Comp. Neurol. 480: 281-298.

Belmonte, M.K., Gomot, M., Baron-Cohen, S., 2010. Visual attention in autism families: "unaffected" sibs share atypical frontal activation. J. Child Psychol. Psychiatry 51, 259–276.

Benavides-Piccione R, Ballesteros-Yanez I, Martinez de Lagran M, Elston G, Estivill X, Fillat C, De Felipe J, Dierssen M. 2004. On dendrites in Down Syndrome and DS murine models: a spiny way to learn. Prog. Neurobiol. 74: 111-126.

Bendz LM, Scates AC. Melatonin Treatment for Insomnia in Pediatric Patients with Attention-Deficit/Hyperactivity Disorder. Ann. Pharmacother. 2010;44(1):185-91.

Beneo Institute. 2009. First Monograph on Isomaltulose Published in Food Chemical Codex. Disponible en: http://www.beneo-group.com/First-monograph-on-isomaltulose-published-in-Food

Benites, L. (1998). Tipos de familia, habilidades sociales y autoestima en un grupo de adolescentes en situación de riesgo. Cultura 16 (12): 191-213

Benites, L., Atención a la diversidad. Guía psicoeducativa para padres y familiares de niños y jóvenes con necesidades educativas especiales. Lima: USMP, 2006

Benitez-Bribiesca L, De la Rosa-Alvarez I, Mansilla-Olivares A. 1999. Dendritic spine pathology in infants with severe protein-calorie malnutrition. Pediatrics 104 (2): 1-6

Bennett FC, mCcLELLAND s, Kriegsmann EA, Andrus LB, Sells CJ. 1983. Vitamin andmineral supplementation in Down's syndrome. Pediatric. 72(5):707-713

Benton D. 2010a. The influence of dietary status on the cognitive performance of children. Mol. Nutr Food Res. 54: 457-470

Benton D. 2010b. Neurodevelopment and neurodegereation: are threre critical stages for nutritional intervention? Nutrition Rev. 68 (Suppl 1):S6-S10

Berkner KL, Runge KW. The physiology of vitamin K nutriture and vitamin K-dependent protein function in atherosclerosis. J Thromb Haemost 2004; 2: 2118–32. Disponible en: http://onlinelibrary.wiley.com/doi/10.1111/j.1538-7836.2004.00968.x/pdf

Bernal Lafuente M, Valdizan JR, García Campayo J. Estudio polisomnográfico nocturno en niños con trastorno por déficit de atención con hiperactividad. Rev Neurol Rev Neurol. 2004;38:103.

Bertalanffy, Ludwing von Teoría General de los Sistemas, México, Fondo de Cultura Económica, Decimoquinta reimpresión, 2003.

Bieberich AA, Morgan SB. 1998. Brief report: Affective expression in children with autism or down syndrome. Journal of Autism and Developmental Disorders 1998;28:333–338. [PubMed: 9711490]

Biederman J, Faraone S, Milberger S, Guite J, Mick I, Chen L, et al. A prospective 4-year follow-up study of attention-deficit hyperactivity and related disorders. Arch Gen Psychiatry. 1996;53:437-46.

Biederman J, Faraone SV, Lapey K. Comorbidity of diagnosis in attention deficit hyperactivity disorder. Child Adolesc Psychiatr Clin N Am. 1992;1:335-60.

Biederman J, Milberger S, Faraone SV, Kiely K, Guite J, Mick E, et al. Family-environment risk factors for attention-deficit hyperactivity disorder. A test of Rutter's indicators of adversity. Arch Gen Psychiatry. 1995;52:464-70.

Biederman J, Thisted RA, Greenhill LL, Ryan ND. Estimation of the association between desipramine and the risk of sudden death in 5- to 14-year-old children. J Clin Psychiatry. 1995;56:87-93.

Billstedt E, Gillberg C, Gillberg C. 2005. Autism after adolescence: Population-based 13- to 22-year followup study of 120 individuals with autism diagnosed in childhood. Journal of Autism and Developmental Disorders 2005;35:351–360. [PubMed: 16119476]

Bittles AH, Bower C, Hussain R, Glasson EJ. 2007. The four ages of Down syndrome. The European Journal of Public Health 2007;17:221–225.

Bittles AH, Glasson EJ. 2004. Clinical, social, and ethical implications of changing life expectancy in Down syndrome. Developmental Medicine and Child Neurology 2004;46:282–286. [PubMed: 15077706]

Blakeborough P, Salter DN, Gurr MI. Zinc binding in cow's milk and human milk. Biochem J 1983; 209:505-12.

Blumer JL, Findling RL, Shih WJ, Soubrane C, Reed MD. Controlled Clinical Trial of Zolpidem for the Treatment of Insomnia Associated With Attention-Deficit/ Hyperactivity Disorder in Children 6 to 17 Years of Age. Pediatrics 2009;123:770-776.

Blunden SL, Milte CM, Sinn N. Diet and sleep in children with attention deficit hyperactivity disorder: Preliminary data in Australian children. J Child Health Care. J Child Health Care. 2011 Mar;15(1):14-24.

Bokkala S, Napalinga K, Pinninti N, Carvalho KS, Valencia I, Legido A, Kothare SV. Correlates of Periodic Limb Movements of Sleep in the Pediatric Population. Pediatr Neurol. 2008;39(1):33-39.

Bokkala S, Napalinga, Pinninti N, Carvalho KS, Valencia I, Legido A, Kothare SV. Correlates of Periodic Limb Movements of Sleep in the Pediatric Population. Pediatr Neurol, 2008;39(1):33-39.

Boure JN, Harris KM. 2008. Balancing structure and function at hippocampal dendritic spines. Ann. Rev. Neurosci. 31:47-67.

Boure JN, Harris KM. 2008. Balancing structure and function at hippocampal dendritic spines. Ann. Rev. Neurosci. 31:47-67.

Bresnahan SM, Anderson JW, Barry RJ. Age-related changes in quantitative EEG in attention-deficitl/hyperactivity disorder. Biol Psychiatry. 1999;46:1690-7.

Brock JW, Prasad C. 1992. Alterations in dendritic spine density in the rat brain associated with protein malnutrition. Brain Res Dev. 66(2): 266-269.

Brockmann PE, Urschitz MS, Noehren A, Sokollik C, Schlaud M, Poets CF. Risk factors and consequences of excessive autonomic activation during sleep in children. Sleep Breath. 2011;15(3):409-16.

Brockmann PE, Urschitz MS, Schlaud M, Poets CF. Primary snoring in school children: prevalence and neurocognitive impairments. Sleep Breath Jan 2011 [Epub ahead of print].

Brown E, editor. Trastornos por déficit de atención y comorbilidad en niños, adolescentes y adultos. Barcelona: Masson; 2003. p. 3-55.

Brown E. Actualización de los trastornos por déficit de atención y sus comorbilidades.

Brown E. Trastorno por déficit de atención con trastornos de sueño. En: Brown E, editor. Trastornos por déficit de atención y comorbilidad en niños, adolescentes y adultos. Barcelona: Masson; 2003. p. 341-62.

Brown FR, Greer MK, Aylward EH, Hunt HH. 1990. Intellectual and adaptive functioning in individuals with Down syndrome in relation to age and environmental placement. Pediatrics. 85: 450-452.

Brown JH, Johnson MH, Patterson SJ, Gilmore R, Longhi E, Karmiloff-Smith A. 2003. Spatial representation and attention in toddlers with Williams syndrome and Down syndrome. Neuropsychol. 41: 1037-1046.

Bruni O, Novelli L, Miano S, Parrino L, Terzano MG, Ferri R. Cyclic alternating pattern: A window into pediatric sleep. Sleep Med. 2010;11(7):628-36.

Bruni O, Novelli L, Miano S, Parrino L, Terzano MG, Ferri R. Cyclic alternating pattern: A window into pediatric sleep. Sleep Med. 2010;11(7):628-36.

Bruni O, Octaviano S, Guidetti V, Romoli M, Innocenzi M, Cortesi F, et al. The Disturbance Scale for Children (SDSC). Construction and validation of an instrument to evaluate sleep disturbances in childhood and adolescence. J Sleep Res. 1996;5: 251-61.5.

Buchs P-A, Muller D. 1996. Induction of long-term potentiation is associated with major ultrastructural changes of activated synapses. Proc. Natl. Acad. Sci. USA. 93: 8040-8045.

Buckley AW, Rodriguez AJ, Jennison K, Buckley J, Thurm A, Sato S, Swedo S. Rapid Eye Movement Sleep Percentage in Children With Autism Compared With Children With Developmental Delay and Typical Development. Arch Pediatr Adolesc. Med. 2010;164(11):1032-1037.

Busby K, Firestone P, Pivik RT. Sleep patterns in hyperkinetic and normal children. Sleep. 1981;4:366-83.

Camfferman D; Kennedy JD; Gold M; Martin AJ; Winwood P; Lushington K. Eczema, sleep, and behavior in children. J Clin Sleep Med 2010;6(6):581-588.

Cantwell DP, Swanson J, Connor DF. Case study: adverse response to clonidine. J Am Acad Child Adolesc Psychiatry. 1997;36:539-44.

Capone G, Goyal ,P, Ares W, Lannigan E. 2006. Neurobehavioral disorders in children, adolescents, and young adults with down syndrome. 2006. Am J Med Gent. 142C:158-176.

Carlesimo GA, Marotta L, Vicari S, 1997. Long-term memory in mental retardation: evidence for a specific impairment in subjects with Down's syndrome. Neuropsychol. 35: 71–79.

Carr J. 2008. The everyday life of adults with Down syndrome. Journal of Applied Research in Intellectual Disabilities 2008;21:389–397.

Carr M, Brodsky L. Sever non obstructive sleep disturbance as an initial presentation of gastroesophageal reflux disease. Int Pediatr Otrohinolaryngol. 1999;51:115-20.

Carvalho SB, Gomes A, Clemente V, Marques M, Pereira AT, Maia B, Soares MJ, Cabral AS, Macedo A, Gozal D, Azevedo MH. Sleep and behavioral/emotional problems in children: A population-based study. Sleep Med. 2009; 10(1): 66-74.

Castellanos FJ, Giedd JN, Berquin PC, Walter JM, Sharp W, Tran T, et al. Quantitative brain magnetic resonance imaging in girls with attentiondeficit/ hyperactivity disorder. Arch Gen Psychiatry. 2001;3:289-95.

Castellanos FJ, Tannock R. Neuroscience of attention-deficit/hyperactivity disorder: the search for endophenotypes. Nature Reviews. 2002;3:617-28.

Chandan, Sen, Savita, Khanna & Sashwati, Roy. (2006). "Tocotrienols: Vitamin E Beyond Tocopherols". Life Sciences Journal. Volume 78, Issue 18, 2088-2098. Disponible en: http://www.ncbi.nlm.nih.gov/pmc/articles/PMC1790869/?tool=pubmed

Chapleau CA, Calfa GD, Lane MC, Albertson AJ, Larimore JL, Kudo S, Armstrong DL, Percy AK, Pozzo-Miller L. 2009. Dendritic spine pathologies in hippocampal pyramidal neurons

from Rett syndrome brain and after expression of Rett-associated MECP2 mutations. Neurobiol Dis. 35(2):219-233.

Chapman RS, Seung H-K, Schwartz SE, Kay-Raining Bird E. 1998. Language skills of children and adolescents with Down syndrome. II. production deficits. J. Speech Lang. Hear Res. 41: 861-873.

Chechlacz M, Gleeson JG. 2003. Is mental retardation a defect of synapse structure and function? Pediatr. Neurol. 29(1):11-17.

Chervin RD, Archbold KH, Dillon JE, Panahi P, Pituch KJ, Dahl RE, et al. Inattention, hyperactivity, and symptoms of sleep disordered breathing. Pediatrics. 2002;109:449-56. 57.

Chervin RD, Archbold KH. Hyperactivity and polysomnographic findings in children evaluated for sleep-disordered breathing. Sleep. 2001;24:313-20.

Chervin RD, Dillon JE, Bassetti C, Ganoczy DA, Pituch KJ. Symptoms of sleep disorders, inattention, and hyperactivity in children. Sleep. 1997;20:1185-92.

Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000;1(1):21-32.

Chervin RD, Ruzicka DL, Hoban TF, Fetterolf JL, Garetz SL, Guire KR, Dillon JE, Felt BT, Hodges EK, Giordani BJ. Esophageal Pressures, Polysomnography, and Neurobehavioral Outcomes of Adenotonsillectomy in Children. Chest. 2012 Feb 2. [Epub ahead of print]

Chiang HL; Shur-Fen Gau S; Ni HC; Chiu YN; Shang CY; Wu YY; Lin; Tai YM; Soong WT. Association between symptoms and subtypes of attention-deficit hyperactivity disorder and sleep problems/disorders. Journal of Sleep Research. 2010;19(4):535-545.

Christianson A, Howson CP, Modell B. 2006. 2006 March of dimes global report on birth defect: The hidden toll of dying and disabled children. White Plains, NY: March of Dimes Birth Defects Foundation. p. 98

Cintra L, Diaz-Cintra S, Galván A, Kemper T, Morgane PJ. 1990. Effects of protein undernutrition on the dentate gyrus in rats of three age groups. Brain Res. 532 (1-2): 271-277.

Clark D, Wilson GN. 2003. Behavioral assessment of children with Down syndrome using the Reiss psychopathology scale. Am. J. Med. Genet. 118: 210–216.

Clarke AR, Barry RJ, McCarthy R, Selikowitz M. EEG analysis in attention-deficit/hyperactivity disorder: a comparative study of two subtypes. Psychiatry Res. 1998;81:19-29.

Cohen AA, Arian A, Harris PA, Byrnes DW, Holzman MD, Sharp KW, et al. Surgical trial investigating nocturnal gastroesophageal reflux and sleep. Surg Edosc. 2003;17:394-400.

Cohen-Zion M, Ancoli-Israel S. Sleep in children with attention-deficit hyperactivity disorder (ADHD): a review of naturalistic and stimulant intervention studies. Sleep Med Rev. 2004;8:379 402.

Comery TA, Harris JB, Willems P J, Oostra BA, Irwin SA, Weiler IJ, Greenough WT. 1997. Abnormal dendritic spines in fragile X knockout mice: Maturation and pruning deficits. Proc. Natl. Acad. Sci. USA. 94: 5401–5404.

Comission of the European Communities. 2005. Comission Decision No 258/97 of the European Parliament and of the Council. Authorization to place Isomaltulose as a Novel Food or Novel Food Ingredient. 25 July 2005. Disponible en: http://eurlex.europa.eu/Notice.do?mode=dbl&lang=en&ihmlang=en&lng1=en,en&lng2=cs,da,de,el,en,es,et,fi,fr,hu,it,lt,lv,nl,pl,pt,sk,sl,sv,&val=405571:cs&page=

Corkum P, Moldofsky H, Hogg-Johnson S, Humphries T, Tannock R. Sleep problems in children with attention-deficit/hyperactivity disorder: impact of subtype, comorbidity, and stimulant medication. J Am Acad Child Adolesc Psychiatry. 1999;38:1285-93.

Corkum P, Panton R, Ironside S, MacPherson M, Williams T. Acute Impact of Immediate Release Methylphenidate Administered Three Times a Day on Sleep in Children with Attention-Deficit/Hyperactivity Disorder. Journal of Pediatric Psychology. 2008;33(4):368-379.

Corkum P, Tannock R, Moldofsky H. Sleep disturbances in children with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 1998;37:637-46.

Coronado Herrera, Martha; Vega y León, Salvador; Gutiérrez Tolentino, Rey; Fernández García, Beatriz & Díaz González, Gilberto (2006). "Los Ácidos Grasos Omega-3 y Omega-6: Nutrición, Bioquímica y Salud". Universidad Nacional Autónoma de México. Revista de Educación Bioquímica, Volumen 25, Número 003, 72-79. Disponible en: http://redalyc.uaemex.mx/src/inicio/ArtPdfRed.jsp?iCve=49025302

Cortese S, Faraone SV, Konofal E, Lecendreux M. Sleep in Children With Attention-Deficit/Hyperactivity Disorder: Meta-Analysis of Subjective and Objective Studies. J Am Acad Child Adolesc Psychiatry. 2009;48(9):894-908
Cortese S, Konofal E, Bernardina BD, Mouren MC, Lecendreux M. Sleep disturbances and serum ferritin levels in children with attention-deficit/hyperactivity disorder. Eur Child Adolesc Psychiatry. 2009;18(7):393-9.

Cortese S, Konofal E, Lecendreux M. Alertness and feeding behaviors in ADHD: does the hypocretin/orexin system play a role? Med Hypotheses. 2008;71(5):770-5.

Cortese S, Morcillo Peñalver C. Comorbidity between ADHD and obesity: exploring shared mechanisms and clinical implications. Postgrad Med. 2010;122(5):88-96.

Cortese S, Vincenzi B. Obesity and ADHD: Clinical and Neurobiological Implications. Curr Top Behav Neurosci. 2012;9:199-218.

Cortesi F, Giannotti F, Ivanenko A, Johnson K. Sleep in children with autistic spectrum disorder. Sleep Med. 2010;11(7):659-64.

Cotton S, Richdale A. 2006. Brief report: Parental descriptions of sleep problems in children with autism, Down syndrome, and Prader-Willi syndrome. Research in Developmental Disabilities 2006;27:151–161. [PubMed: 15975763]

Courchesne, E., Pierce, K., 2005. Why the frontal cortex in autism might be talking only to itself: local over-connectivity but long-distance disconnection. Curr. Opin. Neurobiol. 15, 225–230.

Cruz-Martín A, Crespo M, Portera-Cailliau C. 2010. Delayed stabilization of dendritic spines in fragile X mice. J. Neurosci. 30(23):7793-7803.

Cunnane, Stepehn C.; Hamadeh, Mazen J.; Liede, Andrea C.; Thompson, Lilian U.; Wolever, Thomas MS. & Jenkins, David JA. (1995). "Nutritional Attributes of Traditional Flaxseed in Healthy Young Adults". American Journal of Clinical Nutrition. Volume 61, Number 1, 62 – 68. Disponible en: http://www.ajcn.org/content/61/1/62.full.pdf+html

Curcio G, Ferrara M, De Gennaro L. Sleep loss, learning capacity and academic performance. Sleep Med Rev. 2006;10(5):323-37

Dahl RE, Holttum J, Trubnik L. A clinical picture of child and adolescent narcolepsy. J Am Acad Child Adolesc Psychiatry. 1994;33:834-41.

Dahl RE. Regulation of sleep and arousal: development and psychopathology. Dev Psychopathol. 1996;8:3-27.

Darios, Frédéric & Davletov, Bazbek. (2006). "Omega-3 and Omega-6 Fatty Acids Stimulate Cell Membrane Expansion by Acting on Syntaxin 3". Nautre, International Weekly Journal of Science, Volume 440, 813-817

Daun JK, Przybylski R. 2000. Environmental effects on the composition of four Canadian flax cultivars. Proc. Flax Inst. 58: 80-91.

Davidson LA, Lönnerdal B. Fe saturation and proteolysis of human lactoferrin: effect on brush border receptor mediated uptake of Fe2+ and Mn2+. Am J Physiol 1989; 257:G930-G934.

Dawson G, Meltzoff AN, Osterling J, Rinaldi J, Brown E. Children with autism fail to orient to naturally occurring social stimuli. Journal of Autism and Developmental Disorders 1998;28:479–485. [PubMed: 9932234]

Day HD, Abmayr SB. Parent reports of sleep disturbances in stimulant medicated children with attention-deficit/hyperactivity disorder. J Clin Psychol. 1998;54:701-16.

De Rubens Figueroa J, del Pozzo Magaña B, Pablos Hach JL, Calderón Jiménez C, Castrejón Urbina R. 2003. Malformaciones cardiacas en niños con síndrome de Down. Rev Esp Cardiol. 56:894-899.

DeFelipe J. 2006. Brain plasticity and mental processes: Cajal again. Nat. Rev. Neurosci. 7: 811-817.

Devenny DA, Silverman WP, Hill AL, Jenkins E, Sersen EA, Wisniewski KE. 1996. Normal ageing in adults with Down's syndrome: a longitudinal study. J. Intellect. Disabil. Res. 40:208-221.

Diario de la Salud Medicina Digital. "TDA en México, Un Problema de Salud Pública". 2009. Disponible en: http://www.medicinadigital.com/index.php/salud-mental/13473-TDA-en-mexico-un-problema-de-salud-publica-.html.

Dickstein DL, Kabaso D, Rocher AB, Luebke JI, Wearne SL, Hof PR. 2007. Changes in the structural complexity of the aged brain. Aging Cell. 6:275-284.

Didden R, Sigafoos J, Green VA, Korzilius H, Mouws C, Lancioni GE, O'Reilly MF, Curfs LMG. 2008. Behavioural flexibility in individuals with Angelman syndrome, Down syndrome, non-specific intellectual disability and autism spectrum disorder. Journal of Intellectual Disability Research 2008;52:503–509. [PubMed: 18384537]

Dierssen M, Ortiz-Abalia J, Arque G, Martinez de Lagran M, Fillat C. 2006. Pitfalls and hopes in Down syndrome therapeutic approaches: In the search for evidence-based treatments. Behav. Genet. 36(3):454-468.

Dierssen M, Ramakers GJ. 2006. Dendritic pathology in mental retardation: from molecular genetics to neurobiology. Genes Brain Behav. 5: 48-60.

DiGuiseppi C, Hepburn S, Davis JM, Fidler DJ, Lee NR, Miller L, Ruttenber M, Robinson C. 2010. Screening for autism spectrum disorders in children with Down syndrome: population prevalence and screening test characteristics. J Dev Behav Pediatr. 31(3):181-191.

Dis-Capacidad, Trabajando por la Salud. "Población Down en México". 2010. Disponible en: www.dis-capacidad.com/page/detailsprint.php?id=851

Domínguez L, Pérez-Peñate G. Diagnóstico y tratamiento farmacológico del trastorno por déficit de atención e hiperactividad. Med Clin (Barc). 2003;11:437-38.

Ducros, Veronique; Arnaud, Josaine; Tahiri, Maha; Coudray, Charles; Bornet, Francis; Bouteloup-Demange, Corinne; Brouns, Fred; Rayssiguier, Yves & Roussel, Anne Marie. (2005). "Influence of Short-Chain Fructo-Oligosaccharides (sc-FOS) on Absorption of Cu, Zn and Se in Healthy Postmenopausal Women". Journal of the American College of Nutrition. Vol 24, No 1, 30-37. Disponible en: http://www.jacn.org/content/24/1/30.full.pdf+html

Durmer JS, Dinges DF. Neurocognitive consequences of sleep deprivation. Semin Neurol. 2005;25(1):117-29.

Edal J, Sabbioni E. Vanadium transport across placenta and milk of rats to the fetus and newborn. Biol Trace Ele Res 1989; 22:265-75.

Eisenhower AS, Baker BL, Blacher J. 2005. Preschool children with intellectual disability: Syndrome specificity, behaviour problems, and maternal well-being. Journal of Intellectual Disability Research 2005;49:657–671. [PubMed: 16108983]

Ellis JM, Tan HK, Gilbert RE, Muller DPR, Henley W, Moy R, Pumphrey R, Ani C, Davies A, Logan S. 2008. Supplementation with antioxidants and folinic acid for children with Down's syndrome: randomized controlled trial. Brit. Med. J. 336(7644):594-597.

Esbensen AJ, Seltzer MM, Krauss MW. 2008. Stability and change in health, functional abilities and behavior problems among adults with and without Down syndrome. American Journal on Mental Retardation 2008;113:263–277. [PubMed: 18564887]

Fabiano GA, Pelham WE, Coles EK, et al. A meta-analysis of behavioral treatments for attention deficit/hyperactivity disorder. Clin Psychol Rev. 2009;29:129–140.

Faraone SV, Doyle AE. Genetic influences on attention deficit hyperactivity disorder. Curr Psychiatry Rep. 2000;2:143-6.

Faraone SV, Glatt SJ, Bukstein OG, Lopez FA, Arnold LE, Findling RL. Effects of Once-Daily Oral and Transdermal Methylphenidate on Sleep Behavior of Children With ADHD. J Atten Disord. 2009;12:308-315.

Federal Register number 52783. Vol. 72 No. 179. Monday, September 17th, 2007. Food Labeling; Health Claims; Dietary Noncariogenic Carbohydrate Sweeteners and Dental Caries. Estados Unidos de Norteamérica. Disponible en: http://www.gpo.gov/fdsys/pkg/FR-2007-09-17/pdf/E7-18196.pdf

Feingold BF. Hyperkinesis and learning disabilities linked to artificial food flavors and colors. Am J Nurs. 1975;75:797–803.

Feingold BF. Why Is Your Child Hyperactive? NewYork: Random House; 1975.

Ferber R, Kryger M. Principles and practice of sleep medicine in the child. Philadelphia: WB Saunders; 1995.

Ferrer I, Gullota F. 1990. Down's syndrome and Alzheimer's disease: dendritic spine counts in the hippocampus. Acta Neuropathol. 79: 680-685.

Fiala JC. Spacek J, Harris KM. 2002. Dendritic spine pathology: Cause or consequence of neurological disorders? Brain Res. Rev. 39: 29-54.

Findling RL. Evolution of the treatment of attention-deficit/ hyperactivity disorder in children: a review. Clin Ther. 2008;30:942–957.

Flórez; Jesús. Terapias farmacológicas y suplementos nutritivos para las personas con síndrome de down. Facultad de Medicina, Universidad de Cantabria. Santander. http://www.down21.org/salud/terapias/terapia\_farma.htm

Food and Agriculture Organization of the United Nations & World Health Organization (2001). Report of a Joint FAO/WHO Expert Consultation on Evaluation of Health and Nutritional Properties of Probiotics in Food Including Powder Milk with Live Lactic Acid Bacteria.

Córdoba, Argentina.

http://www.who.int/foodsafety/publications/fs\_management/en/probiotics.pdf

Food and Drug Administration. Appendix F: Calculate the Percent Daily Value for the Appropriate Nutrients. Estados Unidos de Norteamérica. Disponible en: http://www.fda.gov/Food/GuidanceComplianceRegulatoryInformation/GuidanceDocume nts/FoodLabelingNutrition/FoodLabelingGuide/ucm064928.htm

Food and Drug Administration. CFSAN/Office of Premarket Approval. Agency Response Letter GRAS Notice GRN 000052.Estados Unidos de Norteamérica. 30 de Enero 2001. Disponible en:

http://www.fda.gov/Food/FoodIngredientsPackaging/GenerallyRecognizedasSafeGRAS/GRASListings/ucm153729.htm

Food and Drug Administration. CFSAN/Office of Premarket Approval. Agency Response Letter GRAS Notice GRN 000184. March 20th 2006. Disponible en: http://www.accessdata.fda.gov/scripts/fcn/gras\_notices/grn000184.pdf

Frazer A, Gerhardt GA, Daws LC. New views of biogenic amine transporter function: implications for neuropsychopharmacology. Int J Neuropsychopharmacol. 1999;2:305-20.

Frohlich TE, Lanphear BP, Epstein JN, et al. Prevalence, recognition, and treatment of attention deficit/hyperactivity disorder in a national sample of US children. Arch Pediatr Adolesc Med. 2007;161:857–864.

Fukaya, Taisuke; Gondaira, Takumi; Kashiyae, Yasuto; Kotani, Susumu; Ishikura, Yoshiyuki; Fujikawa, Shigeaki; Kiso Yoshinobu & Sakakibara, Manabu. (2005). "Arachidonic Acid Preserves Hippocampal Neuron Membrane Fluidity in Senescent Rats". Neurobiology of Aging, Volume 28, Issue 8, 1179-1186.

Gagliano A, Arico I, Calarese T, Condurso R, Germano E, Cedro C, Spina E, Silvestri R. Restless Leg Syndrome in ADHD children: Levetiracetam as a reasonable therapeutic option. Brain Dev. 2011;33(6):480-6.

Gail Williams P, Sears LL, Allard A. Sleep problems in children with autism. J Sleep Res. 2004;13(3):265-8.

Galaburda AM, Wang PP, Bellusi U, Rossen M. 1994. Cytoarchitectonic anomalies in genetically based disorders: Williams syndrome. Neuroreport. 5(7): 753-757.

Galland BC, Tripp EG, Gray A, Taylor BJ. Apnea-hypopnea indices and snoring in children diagnosed with ADHD: a matched case-control study. Sleep Breath. 2011;15(3):455-62.

Galland BC, Tripp EG, Taylor BJ. The sleep of children with attention deficit hyperactivity disorder on and off methylphenidate: a matched case-control study. J Sleep Res. 2010;19(2):366-73.

Gao X, Lyall K, Palacios N, Walters AS, Ascherio A. RLS in middle aged woman and attention deficit/hyperactivity disorder in their Offspring. Sleep Medicine. 2011;12:89-91.

Garcia-Lopez P, Garcia-Marin V, Freire M. 2007. The discovery of dendritic spines by Cajal in 1888 and its relevance in the present neuroscience. Prog. Neurobiol. 83: 110-130.

Garcia-Ruiz M, Diaz-Cintra S, Cintra L, Corkidi G. 1993. Effect of protein malnutrition on CA3 hippocampal piramidal cells in rats of three ages. Brain Res. 625(2):203-212.

Gau SS, Chiang HL. Sleep problems and disorders among adolescents with persistent and subthreshold attention-deficit/hyperactivity disorders. Sleep. 2009;32(5):671-9.

Gaub M, Carlson CL. Gender differences in ADHD: a meta-analysis and critical review. J Am Acad Child Adolesc Psychiatry. 1997;36:1036-45.

Gershon Michel D. The Second Brain. New York, NY, Quill William Morrow and Company, Inc. Second Edition. 2005.

Gershon, Michael D. (1999). "The Second Brain: A Groundbreaking New Understanding of Nervous Disorders of the Stomach and Intestine". New York, NY, Quill William Morrow and Company, Inc. Second Edition. 2005.

Geschwind, D.H., Levitt, P., 2007. Autism spectrum disorders: developmental disconnection syndromes. Curr. Opin. Neurobiol. 17, 103–111.

GHM van den Heuvel, Ellen; Muys, Theo; van Dokkum, Wim & Schaafsma, Gertjan. (1999). "Oligofructose Stimulates Calcium Absorption in Adolescents". The American Journal of Clinical Nutrition. Vol 69, No 3, 544-548. Disponible en: http://www.ajcn.org/content/69/3/544.full.pdf+html

Giannotti F, Cortesi F, Cerquiglini A, Vagnoni C, Valente D. Sleep in children with autism with and without autistic regression. J Sleep Res. 2011;20(2):338-47.

Giblin JM, Strobel AL. Effect of Lisdexamfetamine Dimesylate on Sleep in Children With ADHD. J Atten Disord. 2011;15:491-498.

Golan N, Shahar E, Ravid S, Pillar G. Sleep disorders and daytime sleepiness in children with attention-deficit/hyperactive disorder. Sleep. 2004;27:261-6.

Golden JA, Hyman BT. 1994. Development of the superior temporal neocortex is anomalous in trisomy 21. J. Neuropathol. Exp. Neurol. 53: 513-520.

Goldman SE, Surdyka K, Cuevas R, Adkins K, Wang L, Malow BA. Defining the sleep phenotype in children with autism. Dev Neuropsychol. 2009;34(5):560-73.

Goodlin-Jones BL, Sitnick SL, Tang K, Liu J, Anders TF. The children's sleep habits questionnaire in toddlers and preschool children. J Dev Behav Pediatr. 2008; 29(2): 82-88.

Goodlin-Jones BL, Tang K, Liu J, Anders TF. Sleep problems, sleepiness and daytime behavior in preschool-age children. J Child Psychol Psychiatry 2009;50(12):1532-40.

Goraya JS, Cruz M, Valencia I, Kaleyias J, Khurana DS, Hardison HH, Marks H, Legido A, Kothare SV. Sleep study abnormalities in children with attention deficit hyperactivity disorder. Pediatr Neurol, 2009; 40(1): 42-6.

Gottlieb DJ, Vezina RM, Chase C, Lesko SM, Heeren TC, Weese-Mayer DE, et al. Symptoms of sleep-disordered breathing in 5-year-old children are associated with sleepiness and problem behaviours. Pediatrics. 2003;112:870-7.

Gozal D, Kheirandish-Gozal L. Neurocognitive and behavioral morbidity in children with sleep disorders. Curr Opin Pulm Med. 2007 Nov;13(6):505-9.

Gozal D. Sleep-disordered breathing and school performance in children. Pediatrics. 1998;102:616-20.

Greenhill L, Puig-Antich J, Goetz R, Hanlon C, Davies M. Sleep architecture and REM sleep measures in prepubertal children with attention deficit disorder with hyperactivity. Sleep. 1983;6:91-101.

Gruber R, Sadeh A, Raviv A. Inestability of sleep patterns in children with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2000;39:495-501.

Gruber R, Sadeh A. Sleep and neurobehavioral functioning in boys with attention-deficit/hyperactivity disorder and no reported breathing problems. Sleep. 2004;27:267-73.

Gruber R; Wiebe S; Montecalvo L; Brunetti B; Amsel R; Carrier J. Impact of sleep restriction on neurobehavioral functioning of children with attention deficit hyperactivity disorder. Sleep. 2011;34(3):315-323.

Guilleminault C, Winkle R, Korobkin R, Simmons B. Children and nocturnal snoring-evaluation of the effects of sleep related respiratory resistive load and daytime functioning. Eur J Pediatr. 1982;139:165 71.

Gundappa G, Desiraju T. 1988. Deviations in brain development of F2 generation on caloric undernutrition and scope of their prevention by rehabilitation: alterations in dendritic spine production and pruning of pyramidal neurons of lower laminae of motor cortex and visual cortex. Brain Res. 456(2):205-223.

Haboud H. New therapeutic possibilities in mongolism, suggestions for specific treatments. Arzeneimittel Forschung, 9:211-228, 1955.

Hagerman RJ, Falkenstein AR. An association between recurrent otitis media in infancy and later hyperactivity. Clin Pediatr. 1987;26:253-7.

Hansen B, Skirbekk B, Oerbeck B, Richter J, Kristensen H. Comparison of sleep problems in children with anxiety and attention deficit/hyperactivity disorders. European Child & Adolescent Psychiatry. 2011;20(6):321-30.

Harrell RF. Can nutritional supplements help mentally retarded children? An exploratory study. Proceedings of the National Academy of Sciences USA 78:574-578, 1981.

Hering E, Epstein R, Elroy S, Iancu DR, Zelnik N. Sleep patterns in autistic children. J Autism Dev Disord. 1999;29(2):143-7.

Hering H, Sheng M. 2001. Dendritic spines: structure, dynamics and regulation. Nat. Rev. Neurosci. 2: 880-888.

Herman, Janice R. "Protein and the Body" División de Ciencias de la Agricultura y Recursos Naturales. Universidad Estatal de Oklahoma. Disponible en: http://pods.dasnr.okstate.edu/docushare/dsweb/Get/Document-2473/T-3163web2011.pdf

Hodapp RM, Ewans DE, Gray FL. 1999. Intellectual development in children with Down syndrome. En Rondal JA, Perea J, Nadel L (Eds). Down Syndrome: A review of current knowledge. Whurr Publisher, London pp. 124 132.

Hoebert M, van der Heijden KB, van Geijlswijk IM, Smits MG. Long-term follow-up of melatonin treatment in children with ADHD and chronic sleep onset insomnia. J Pineal Res. 2009;47(1):1-7.

Holland, AJ. 1999. Down's syndrome. In: Janicki, MP.; Dalton, AJP., editors. Dementia and Aging Adults with Intellectual Disability: A Handbook. Philadelphia, PA: Taylor & Francis; 1999. p. 183-197.

Hoppes K, Harris SL. 1990. Perceptions of child attachment and maternal gratification in mothers of children with autism and Down syndrome. Journal of Clinical Child Psychology 1990;19:365–370.

Howlin P, Goode S, Hutton J, Rutter M. 2004. Adult outcome for children with autism. Journal of Child Psychology and Psychiatry 2004;45:212–229. [PubMed: 14982237]

http://www.inei.gob.pe/biblioinei.asp

Hunter, J.W., Mullen, G.P., McManus, J.R., Heatherly, J.M., Duke, A., Rand, J.B., 2010. Neuroligin deficient mutants of C. elegans have sensory processing deficits and are hypersensitive to oxidative stress and mercury toxicity. Dis. Model Mech 3,366–376.

Hvolby A, Jorgensen J, Bilenberg N. Actigraphic and Parental Reports of Sleep Difficulties in Children With Attention-Deficit/Hyperactivity Disorder. Arch Pediatr Adolesc Med. 2008;162(4):323-329.

Hvolby A, Jorgensen J, Bilenberg N. Parental rating of sleep in children with attention deficit/hyperactivity disorder. Eur Child Adolesc Psychiatry. 2009;18(7):429-38.

Hyo-Won K, In-Young Y, Soo-Churl C, Boong-Nyun K, Seockhoon C, Hyewon L, chi-Won K, sung-Kun P, Hee Jeong Y. The effect of OROS methylphenidate on the sleep of children with attention-deficit/hyperactivity disorder. Int Clin Psycopharmacol. 2010;25(2):107-15.

Ingram S, Hechtman L, Mrgerstern G. Outcomes issues in ADHD: adolescent and adult long-term outcomes. Ment Retard Dev Disabil Res Rev. 1999;5:243-50. 72. 73.

Instituto Nacional de Estadística e informática (2002) Qué es la teoría general de sistemas [en línea] Colección cultura informática,

Jacobs, Eric J. & White, Emily. (1998). "Constipation, Laxative Use, and Colon Cancer among Midel-Aged Adults". Epidemiology Journal. Volume 9, Issue 9, 385-391.

Jamain, S., Quach, H., Betancur, C., Råstam, M., Colineaux, C., Gillberg, I.C., Soderstrom, H., Giros, B., Leboyer, M., Gillberg, C., Bourgeron, T., 2003. Mutations of the X linked genes encoding neuroligins NLGN3 and NLGN4 are associated with autism. Nat. Genet. 34, 27–29.

Jensen PS, Mrazek D, Knapp PK, Steinberg L, Pfeffer C, Schowalter J, et al. Evolution and revolution in child psychiatry: ADHD as a disorder of adaptation. J Am Acad Child Adolesc Psychiatry. 1997;36:1672-9.

Ji NY, Capone GT, Kaufmann WE. 2011. Autism spectrum disorders in Down syndrome: cluster analysis of aberrant behavior checklis data supports diagnosis. J Intellec Dis Res. 55 (11): 10064-1077.

Johnstone SJ, Tardif HP, Barry RJ, Sands T. Nasal bilevel positive airway pressure therapy in children with a sleep-related breathing disorder and attention-deficit hyperactivity disorder: effects on electrophysiological measures of brain function. Sleep Medicine. 2001;2:407-16.

Kado-Oka, Y.; Fujiwara, S. & Hirota, T. (1991). "Effects of Bifidobacteria Cells on Mitogenic Response of Splenocytes and Several Functions of Phagocytes". Milchwissenschaft, Vol 46, 626-630.

Kan, Inna; Melamed, Eldad; Offen, Daniel & Green, Pnina. (2006). "Docosahexaenoic Acid and Arachidonic Acid are Fundamental Supplements for the Induction of Neuronal Differentiation". Journal of Lipid Research. Volume 48, 513-517. Disponible en: http://www.jlr.org/content/48/3/513.full.pdf+html

Kaplan HI, Sadock BJ. Sinopsis de psiquiatría-ciencias de la conducta. 8.a ed. Buenos Aires: Médica Panamericana; 1999.

Kasari C, Hodapp R. ¿Es diferente el síndrome de Down? Datos de estudios sociales y familiares. España, Revista Síndrome Down, 1997.

Kasari C, Sigman M. 1997. Linking parental perceptions to interactions in young children with autism. Journal of Autism and Developmental Disorders 1997;27:39–57. [PubMed: 9018581]

Kasetsart J. (2000). "Production of β-Fructofuranosidasa from Aspergillus niger ATCC 20611". National Science Journal. Vol 34, 378-386. Disponible en: http://pindex.ku.ac.th/file\_research/Product378-386.pdf

Kasetsart J. (2000). "Production of β-Fructofuranosidase from Aspergillus niger ATCC 20611". National Science Journal. Vol 34, 378-386. Disponible en: http://pindex.ku.ac.th/file\_research/Product378-386.pdf

Kaufmann WE, Moser HW. 2000. Dendritic anomalies in disorders associated with mental retardation. Cereb. Cortex. 10:981-991.

Kawai, K., Okuda, Y., Yamashita, K. 1985. Changes in blood glucose and insulin after an oral palatinose administration in normal subjects. Edocrinolgia Japonica 32, 933-936. Disponible en: https://www.jstage.jst.go.jp/article/endocrj1954/32/6/32\_6\_933/\_article

Kemper TL, Pasquier DA, Drazen S. 1978. Brain Res Bull. 3(5):443-450

Kent JD, Blader JC, Koplewicz HS, Abikoff H, Foley CA. Effects of late-afternoon methylfenidate administration on behaviour and sleep in attention-deficit hyperactivity disorder. Pediatrics. 1995;96:320-5.

Kim JK, Lee JH, Lee SH, Hong SC, Cho JH. School performance and behavior of Korean elementary school students with sleep-disordered breathing. Ann Otol Rhinol Laryngol. 2011;120(4):268-72.

Kim SJ, Lee YJ, Cho SJ, Cho I-H, Lim W, Lim W. Relationship Between Weekend Catch-up Sleep and Poor Performance on Attention Tasks in Korean Adolescents. Arch Pediatr Adolesc Med. 2011;165(9):806-812.

Kirk V, Kahn A, Brouillette RT. Diagnostic approach to obstructive sleep apnea in children. Sleep Med. 1998;2:255-69.

Kirkman Labs. "Buffered Magnesium Glycinate Powder - Bio-Max Series - New, Improved Formula". Disponible en: http://kirkmanlabs.com/ProductKirkman/327/1/Buffered%20Magnesium%20Glycinate%C

2%AE%20Powder%20-%20Bio-Max%20Series%20-%20New,%20Improved%20Formula/

Kirkman Labs. "Products by Function". Disponible en: http://kirkmanlabs.com/ProductsByFunctionIndex.aspx

Kirov R, Pillar G, Rothenberger A. REM-sleep changes in children with attention-deficit/hyperactivity disorder: methodologic and neurobiologic considerations. Sleep. 2004;27:1215.

Knobloch M, Mansuy IM. 2008. Dendritic spine loss and synaptic alterations in Alzheimer's disease. Mol. Neurobiol. 37:73-82.

Kohwi, Yoshinori; Hashimito, Yoshiyuki & Tamura, Zenzo. (1982). "Antitumor and Immunological Adjuvant Effect of Bifidobacterium Infantis in Mice". Departamento de Química de la Higiene del Instituto Farmacéutico, Universidad de Tohoku. Departamento de Farmacéutica de la Escuela de Medicina de la Univesidad de Tokio. Bifidobacteria Microflora, Vol 1, 61-68. Disponible en: https://www.jstage.jst.go.jp/article/bifidus1982/1/1/1\_1\_61/\_pdf

König, Daniel; Theis, Stephan, Kozianowski, Gunhild & Berg, Aloys. (2011). "Postprandial Substrate Use in Overweight Subjects With The Metabolic Syndrome After Isomaltulose (Palatinose) Ingestion". Departament of Rehabilitation, Prevention and Sports Medicine, Center for Internal Medicine, University Hospital Feiburg. Beneo. Germany. http://www.sciencedirect.com/science/article/pii/S0899900711003613

Konofal E, Lecendreux M, Bouvard MP, Mouren-Simeoni MC. High levels of nocturnal activity in children with attention-deficit hyperactivity disorder: a video analysis. Psychiatry Clin Neurosci. 2001;55:97-103.

Konofal E, Lecendreux M, Cortese S. Sleep and ADHD. Sleep Med. 2010;11(7):652-8.

Krakowiak P, Goodlin-Jones B, Hertz-Piccioto I, LA Croen LA, Hansen RL. Sleep problems in children with autism spectrum disorders, developmental delays, and typical development: a population-based study. J Sleep Res. 2008; 17(2): 197-206.

Kune, Gabriel A.; Kune, Susan; Field, Barry & Watson, Lyndsey F. (1998). "The Role of Chronic Constipation, Diarrhea, and Laxative Use in the Etiology of Large Bowel Cancer. Data from the Melbourne Colorectal Cancer Study". Diseases of the Colon & Rectum, Volume 31, Number 7, 507-512

Kuperman S, Johnson B, Arndt S, Lindgren S, Wolraich M. Quantitative EEG differences in a nonclinical sample of children with ADHD and undifferentiated ADD. J Am Acad Child Adolesc Psychiatry. 1996;8:1009-17.

Laberge L, Tremblay RE, Vitaro F, Montplaisir J. Development of parasomnias from childhood to early adolescence. Pediatrics. 2000;106(1 Pt 1):67-74.

Landau YE, Bar-Yishay O, Greenberg-Dotan S, Goldbart AD, Tarasiuk A, Tal A. Impaired behavioral and neurocognitive function in preschool children with obstructive sleep apnea. Pediatr Pulmonol. 2012;47(2):180-8.

LeBourgeois MK, Avis K, Mixon M, Olmi J, Harsh J. Snoring, sleep quality and sleepiness across attention-deficit hyperactivity disorder subtypes. Sleep. 2004;27:520-5. 58.

Lecendreux M, Konofal E, Bouvard M, Falissard B, Mouren-Simeoni MC. Sleep and alertness in children with ADHD. J Child Psychol Psychiatry. 2000;41:803-12. 45. 46.

Leu RM, Beyderman L, Botzolakis EJ, Surdyka K, Wang L, Malow BA. Relation of Melatonin to Sleep Architecture in Children with Autism. J Autism Dev Disord. 2011;41(4):427-33.

Levay, Peter F; Viljoen, Margaretha (1995). Haematologica Journal. Volume 80, Issue 3, Pages 252-267: Lactoferrin: A General Review. Departament of Phisiology, University of Pretoria, South Africa. Disponible en: http://www.haematologica.org/content/80/3/252.long

Li JM, Hu JT, Luo XM, Cai YM, Liu JM. [Correlation of snoring with attention deficit and hyperactivity-impulsivity in school age children from Changsha City. Zhongguo Dang Dai Er Ke Za Zhi. 2009;11(7):562 5.

Li S, Jin X, Yan C, Wu S, Jiang F, Shen X. Sleep Problems in Chinese School-Aged Children with a Parent-Reported History of ADHD. J Atten Disord. 2009;13:18-26.

Li Z, Sheng M. 2003. Some assembly required: the development of neuronal synapses. Nat. Mol. Cell Biol. 4: 833-841.

Lichstein, Herman C.; Gunsalus, I.C. & Umbreit, W.W. (1945). "Function of the Vitamin B6 Group: Pyridoxal Phosphate (Codecarboxylase) in Transamination". Journal of Biological Chemistry. Volume 161, 311 - 320.

Lina, B.A.R.; Jonker, D.; Kozianowski, G. (2002). "Isomaltulose (Palatinose): A review of biological and toxicological studies". Food and Chemical Toxicology 40 (10): 1375–81. http://www.sciencedirect.com/science/article/pii/S0278691502001059

Lintas, C., Persico, A.M., 2009. Autistic phenotypes and genetic testing: state-of-the-art for the clinical geneticist. J. Med. Genet. 46, 1–8.

Lintas, Carla Lintas; Sacco, Roberto; Persico, Antonio M. Genome-wide expression studies in Autism spectrum disorder, Rett syndrome, and Down syndrome. Neurobiology of Disease

Volume 45, Issue 1, January 2012, Pages 57–68 Assessment of Gene Expression in Neuropsychiatric Disease. Laboratory of Molecular Psychiatry and Neurogenetics, University "Campus Bio-Medico", Rome, Italy. Department of Experimental Neurosciences, I.R.C.C.S. "Fondazione Santa Lucia", Rome, Italy.

Lipp HP, Wolfer DP.1998. Genetically modified mice and cognition. Curr. Opin. Neurobiol. 8:272-280.

Lockrow J, Prakasam A, Huang P, Bimonte-Nelson H, Sambamurti K, Granholm AC. 2009. Cholinerrgic degeneration and memory loss delayed by vitamin E in Down syndrome mouse model. Exp. Neurol. 216 (2):278-289.

Loot I, Dierssen M. 2010. Cognitive deficits and associated neurological complications in individuas with Down's syndrome. Lancet Neurol. 9: 623-33.

Lott IT, Head E. 2005. Alzheimer disease and Down syndrome: factor in pathogenesis. Neurobiol. Aging. 26:383-389.

Luckasson, R.; Borthwick-Duffy, S.; Buntinx, WHE.; Coulter, DL.; Craig, EM.; Reeve, A.; Schalock, RL.; Snell, ME.; Spitalnik, DM.; Spreat, S.; Tassé, MJ. 2002. Mental retardation: Definition, classification, and systems of supports. 10th. Washington, DC: American Association on Mental Retardation; 2002.

Maatta T, Tervo-Maatta T, Taanila A, Kaski M, Iivanainen M. 2006. Mental Health, behavior and intellectual abilities of people with Down syndrome. Down Synd Res Pract. 11 (1):37-43

Mahoney FE, Barthel DW. Functional evaluation: The Barthel Index. Maryland State Medical Journal 1965;14:61–65. [PubMed: 14258950]

Malow BA, Crowe C, Henderson L, McGrew SG, Wang L, Song Y, Stone WL. A Sleep Habits Questionnaire for Children With Autism Spectrum Disorders. J Child Neurol, 2009; 24: 19 - 24.

Malow BA, Marzec ML, McGrew SG, Wang L, Henderson LM, Stone WL. Characterizing sleep in children with autism spectrum disorders: a multidimensional approach. Sleep. 2006;29(12):1563-71.

Mann CA, Lubar JF, Zimmerman AW, Miller CA, Muenchen RA. Quantitative analysis of EEG in boys with attention-deficit/hyperactivity disorder: controlled study with clinical implications. Pediatr Neurol. 1992;8:30-6.

Manocha, M; Shajib, MS; Rahman, MM; Wang, H; Rengasamy, P; Bugonovic, M; Jordana, M; Mayer, L & Khan, I. (2012). "IL-13-Mediated Immunological Control of Enterochormafiin Cell Hyperplasia and Serotonin Production in the Gut". Mucosal Immunology Journal. Nature

Publishing Group. Disponible en: http://www.nature.com/mi/journal/vaop/ncurrent/full/mi201258a.html

Marin-Padilla M. 1972. Structural abnormalities of the cerebral cortex in human chromosomal aberrations: A Golgi study. Brain Res. 44: 625-629.

Marin-Padilla M. 1976. Pyramidal cell abnormalities in the motor cortex of a child with Down's syndrome: A Golgi study. J. Comp. Neurol. 167: 63-81.

Martin HP. 1973. Nutrition: its relationship to children's physical, mental, and emotional development. Am. J. Clil. Nutrit. 26:766-775.

Matsuzaki M, Honkura N, Ellis-Davies GC, Kasai H. (2004) Structural basis of long-term potentiation in single dendritic spines. Nature. 429:761-766.

Matthews Julie, Nourishing Hope for Autism. Healthful Living Media, Third Edition, 2008

Mauro, Terri. The Everything Parents Guide, Sensory Integration Disorder, Avon, MA, Adams Media a division of

Max JE, Fox PT, Lancaster JL, Kochunov P, Mahtews K, Manes FF, et al. Putamen lesions and the development of attention-deficit/hyperactivity symptomatology. J Am Acad Child Adolesc Psychiatry. 2002;41:563-71.

Mayes SD, Calhoun SL, Bixler EO, Vgontzas AN, Mahr F, Hillwig-Garcia J, Elamir B, Edhere-Ekezie L, Parvin M. ADHD Subtypes and Comorbid Anxiety, Depression, and Oppositional-Defiant Disorder: Differences in Sleep Problems. Journal of Pediatric Psychology 2009 34(3):328-337.

McCanless Jaquelyn , MD. Children with Starving Brains. Bramble Books, Fourth Edition. 2009.

McConnell P, Berry M. 1979. The effects of postnatal lead exposure on Purkinje cell dendritic development in the rat. Neuropathol Appl Neurobiol. 5(2):115-132.

McCormick, D. B. Vitamin B6 In: Present Knowledge in Nutrition (Bowman, B. A. and Russell, R. M., eds), 9th edition, vol. 2, p.270. Washington, D.C.: International Life Sciences Institute, 2006.

Melendez-Ferro M, Perez-Costas E, Roberts RC. 2009. A new use for long-term fozen brain tissue: golgi impregnation. J. Neurosci. Meth. 176(2):72-77.

Meléndez-Hevia E, Waddell TG, Cascante M (1996). "The puzzle of the Krebs citric acid cycle: assembling the pieces of chemically feasible reactions, and opportunism in the

design of metabolic pathways during evolution". J. Mol. Evol. 43 (3): 293–303. Disponible en: http://www.ncbi.nlm.nih.gov/pubmed/8703096

Meltzer LJ, Johnson C, Crosette J, Ramos M, Mindell JA. Prevalence of Diagnosed Sleep Disorders in Pediatric Primary Care Practices. Pediatrics. 2010 Jun;125(6):e1410-8. Epub 2010 May 10.

Meltzer LJ, Johnson C, Crosette J, Ramos M, Mindell JA. Prevalence of Diagnosed Sleep Disorders in Pediatric Primary Care Practices. Pediatrics. 2010;125(6):1408-10.

Meng Y, Zhang Y, Tregoubou V, Janus C, Cruz L, Jackson M, Luw Y, MacDonald JF, Wang JY, Falls DL, Jia Z. 2002. Abnormal spines morphology and enhanced LTP in LIMK-1 knockout mice. Neuron. 35(1): 121-133.

Menzies, I.S., 1974. Absorption of intact oligosaccharide in health and disease. Biochemical Society Transactions 2, 1042–1047.

Miano S, Ferri R. Epidemiology and management of insomnia in children with autistic spectrum disorders. Paediatr Drugs 2010;12(2):75-84

Miano S, Paolino MC, Urbano A, Parisi P, Massolo AC, Castaldo R, Villa MP. Neurocognitive assessment and sleep analysis in children with sleep-disordered breathing. Clin Neurophysiol. 2011;122(2):311-9.

Mick E, Biederman J, Faraone SV, Sayer J, Kleinman S. Case-control study of attention-deficit hyperactivity disorder and maternal smoking, alcohol use, and drug use during pregnancy. J Am Acad Child Adolesc Psychiatry. 2002;41:378-85.

Mindell JA, Owens JA. A clinical guide to pediatric sleep: diagnosis and management of sleep problems. Philadelphia: Lippincott Williams & Wilkins; 2003.

Mirre, Juan Carlos (2012). "La Importancia del Segundo Cerebro". Revista Discovery DSalud. Número 147. Marzo 2012. España. Disponible en: http://www.dsalud.com/index.php?pagina=articulo&c=1689

Mitsuoka, T., Hidaka, H. and Eida, T. (1987). Departamento de Ciencias Biomédicas, Facultad de Agricultura, Universiad de Tokio, Effect of fructo-oligosaccharides on intestinal microflora. Molecular Nutrition, Food Research. Vol 31. Issue 5-6. 427-436. Japón. DOI: 10.1002/food.19870310528

http://onlinelibrary.wiley.com/doi/10.1002/food.19870310528/abstract

Molis, Christine; Flourié, Bernard; Ouarné, Françoise; Gailing, Marie-Frédérique; Lartigue, Sylvie; Guibert, Alain; Brnoet, Francis & Galmiche, Jean-Paul. (1996). "Digestion, Excretion and Energy Value of Fructooligosaccharides in Healthy Humans". The Amercian Journal of

Clinical Nutrition. 324-328. Disponible en: http://www.educapalimentos.org/site2/archivos/investigaciones/FOS-1.pdf

Moon J, Chen M, Gandhy SU, Strawderman M, Levitsky DA, Maclean KN, Strupp BJ. 2010. Perinatal Choline supplementation improves cognitive function and emotion regulation in the Ts65Dn mouse model of down syndrome. Behav. Neurosci. 124 (3): 346-361.

Moren, I, Los trastornos por déficit de atención con hiperactividad. En M. Servera (coord), Intervención en los trastornos del comportamiento infantil, Madrid, Pirámide, 2002

Morgane PJ, Austin-LaFrance R, Bronzio J, Tonkiss J, Diaz-Cintra S, Cintra L, Kemper T, Galler JR. 1993. Prenatal malnutrition and development of the brain. Neurosci Biobehav Res. 17 (1):91-128

Morice E, Andreae LC, Cooke SF, Vanes L, Fisher EMC, Tybulewicz VLJ, Bliss TVP. 2008. Preservation of long-term memory and synaptic plasticity despite short-term impairments in the Tc1 mouse model of Down syndrome. Learn. Mem. 15: 492-500.

Morris, Diane H. (2007). Linaza – Una Recopilación Sobre sus Efectos en la Salud y Nutrición. 4ª edición. Consejo Canadiense de la Linaza. Disponible en: http://www.flaxcouncil.ca/spanish/index.jsp?p=primer\_spanish

Morris, Martha Clare; Evans, Denis A,; Tangney Christine C.; Bienias, Julia L.; Wilson, Robert S.; Aggarwal, Neelum T.& Scherr, Paul A. (2005). Relation of the tocopherol forms to incident Alzheimer disease and to cognitive change. The American Journal for Clinical Nutrition. Volume 81, Issue 2, 508-514. Disponible en: http://www.ajcn.org/content/81/2/508.abstract

Naczk, Marian & Shahidi, Fereidoon. (2006). "Phenolics in Cereals, Frutis and Vegetables: Occurrence, Extraction and Analysis". Journal of Pharmaceutical and Biomedical Analysis, Volume 41, Issue 5, 1523-1542.

Nadel L. 2003. Down's syndrome: a genetic disorder in biobehavioral perspective. Genes Brain Behav. 2: 156 166.

Nagasawa, Taro; Kiyosawa, Isao & Kuwahara, Kunisuke. (1972). Journal of Dairy Science. Volume 55, Issue 12, Pages 1651-1659: Amounts of Lactoferrin in Human Colostrum and Milk. Tokyo, Japan. Disponible en: http://download.journals.elsevierhealth.com/pdfs/journals/0022-0302/PIIS0022030272857412.pdf

Nagerl UV, Eberhorn N, Cambridge SB, Bonhoeffer T. 2004. Bidirectional activity-dependent morphological plasticity in hippocampal neurons. Neuron. 44:759-767.

Najib J. The efficacy and safety profile of lisdexamfetamine dimesylate, a prodrug of damphetamine, for the treatment of attention-deficit/hyperactivity disorder in children and adults. Clin Ther. 2008;31:142 176.

Noback CR, Eisenman LM. 1981. Some effects of protein-caorie undernutrition on developing central neurvoussystem of the rat. Anat Rec. 201(1):67-73.

Nováková M, Paclt I, Ptáček R, Kuželová H, Hájek I, Sumová A. Salivary Melatonin Rhythm as a Marker of the Circadian System in Healthy Children and Those With Attention-Deficit/Hyperactivity Disorder. Chronobiology International. 2011;28(7):630-637.

Núñez B. Familia y discapacidad de la vida cotidiana a la teoría, Buenos Aires, Lugar Editorial, 2007.

O´connor, Joseph & McDermott, Ian Introducción al pensamiento sistémico, Madrid, URANO, 1998.

O'Brien LM, Holbrook CR, Mervis CB, Klaus CJ, Bruner JL. Sleep and neurobehavioral characteristics of 5- to 7-year-old children with parentally reported symptoms of attention-deficit/hyperactivity disorder. Pediatrics. 2003;111:554-64.

O'Callaghan FV, Al Mamun A, O'Callaghan M, Clavarino A, Williams GM, Bor W, Heussler Najman J. The link between sleep problems in infancy and early childhood and attention problems at 5 and 14years: Evidence from a birth cohort study. Early Hum Dev. 2010;86(7):419-24.

O'Doherty, A., Ruf, S., Mulligan, C., Hildreth, V., Errington, M.L., Cooke, S., Sesay, A., Modino, S., Vanes, L., Hernandez, D., et al. 2005. An aneuploid mouse strain carrying human chromosome 21 with Down syndrome phenotypes. Science 309: 2033–2037

O'Neill DK, Happé FGE.2000. Noticing and commenting on what's new: Differences and similarities among 22-month-old typically developing children, children with Down syndrome and children with autism. Developmental Science 2000;3:457–478.

Oner O, Oner P, Bozkurt OH, et al. Effects of zinc and ferritin levels on parent and teacher reported symptoms scores in attention deficit hyperactivity disorder. Child Psychiatry Hum Dev. 2010;41:441-447.

Owens JA, Dalzell V. Use of the 'BEARS' sleep screening tool in a pediatric residents' continuity clinic: a pilot study. Sleep Medicine. 2005; 6(1):63-9.

Owens JA, Maxim R, Nobile C, McGuinn M, Msall M. Parental and self report of sleep in children with attention-deficit/hyperactivity disorder. Arch Pediatr Adolesc Med. 2000;154:549-55.

Owens JA, Mehlenbeck R, Lee J, King MM. Effect of Weight, Sleep Duration, and Comorbid Sleep Disorders on Behavioral Outcomes in Children With Sleep-Disordered Breathing. Arch Pediatr Adolesc Med. 2008;162(4):313-321.

Owens JA, Mindell JA. Pediatric insomnia. Pediatr Clin North Am. 2011 Jun;58(3):555-69.

Owens JA, Rosen CL, Mindell JA, Kirchner HL. Use of pharmacotherapy for insomnia in child psychiatry practice: A national survey. Sleep Med. 2010; 11(7): 692-700.

Owens JA, Rosen CL, Mindell JA. Medication use in the treatment of pediatric insomnia: results of a survey of community-based pediatricians. Pediatrics. 2003;111:628-

Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000;23(8):1043-51.

Patterson D, Costa ACS. 2005. Down syndrome and genetics-a case of linked histories. Nat. Rev. Gent. 6: 137 147.

Patzold LM, Richdale AL, Tonge BJ. An investigation into sleep characteristics of children with autism and Asperger's Disorder. J Paediatr Child Health. 1998;34(6):528-33.

Pelsser LM, Frankena K, Buitelaar JK, Rommelse NN. Effects of food on physical and sleep complaints in children with ADHD: a randomised controlled pilot study. Eur J Pediatr. 2010;169(9):1129-38.

Pennnington BF, Moon J, Edgin J, Stedron J, Nadel L. 2003. The neuropsychology of Down syndrome: evidence for hippocampal dysfunction. Child Develop. 74: 75-93.

Penzes P, Cahill ME, Jones KA, VanLeeuwen J-C, Woolfrey KM. 2011. Dendritic spine pathology in neuropsychiatric disorders. Nat. Neurosci. 14: 3: 285-293.

Periódico La Jornada. La Jornada en la Ciencia. "Hay 37 mil niños Autistas en México". 2010. Disponible en: http://ciencias.jornada.com.mx/noticias/hay-37-mil-ninos-autistas-en-mexico

Picchietti DL, England SJ, Walters AS, Willis K, Verrico T. Periodic limb movement disorder and restless legs syndrome in children with attention- deficit hyperactivity disorder. J Child Neurol. 1998;13:588-94.

Picchietti DL, Walters AS. Moderate to severe periodic limb movement disorder in childhood and adolescence. Sleep. 1999;22:297-300.

Picchietti DL, Walters AS. Restless legs syndrome and periodic limb movement disorder in children and adolescents: comorbidity with attentiondeficit hyperactivity disorder. Child Adolesc Psychiatr Clin N Am. 1996; 5:729-40.

Picchietti MA; Picchietti DL; England SJ; Walters AS; Couvadelli BV; Lewin DS; Hening W. Children show individual night-to-night variability of periodic limb movements in sleep. Sleep 2009;32(4):530-535.

Pinter, J.D., Eliez, S., Schmitt, J.E., Capone, G.T., Reiss, A.L., 2001. Neuroanatomy of Down's syndrome: a high-resolution study. Am. J. Psychiatry. 58, 1659–1665

Pope AM, Tarlov AR. 1991. Disability in America: toward a National Agenda for Prevention. Washington, DC. National Academic.

Prehn-Kristensen A, Göder R, Fischer J, Wilhelm I, Seeck-Hirschner M, Aldenhoff J, Baving L. Reduced sleep-associated consolidation of declarative memory in attention-deficit/hyperactivity disorder. Sleep Med. 2011 Aug;12(7):672-9.

Prehn-Kristensen A, Molzow I, Munz M, Wilhelm I, Müller K, Freytag D, Wiesner CD, Baving L. Sleep restores daytime deficits in procedural memory in children with attention-deficit/hyperactivity disorder. Res Dev Disabil. 2011;32(6):2480-8.

Prihodova I, Paclt I, Kemlink D, Skibova J, Ptacek R, Nevsimalova S. Sleep disorders and daytime sleepiness in children with attention-deficit/hyperactivity disorder: A two-night polysomnographic study with a multiple sleep latency test. Sleep Med . 2010;11(9):922-8.

Pueschel, Siegfried M, Pueschel, Jeanette K. Biomedical Concerns in Persons with Down Syndrome .Baltimore, Maryland, Paul H. Brookes Publishing Co. 1992

Pullen SJ; Wall CA; Angstman ER; Munitz GE; Kotagal S. Psychiatric comorbidity in children and adolescents with restless legs syndrome: a retrospective study. J Clin Sleep Med. 2011;7(6):587-596.

Pulsifer, MB. 1996. The neuropsychology of mental retardation. J. Int. Neuropsychol. Soc. 2: 159–176.

Purpura DP. 1974. Dendritic spine "dyagenesis" and mental retardation. Science. 186:1126-1128.

Ramos MJ, Vela A, Espinar J, Kales S. Hypnopolygraphic alterations in attention deficit disorder (ADD) children. Int J Neurosci. 1990;53:87-101.

Rapp Doris, M.D. Is this your Child? New York, NY, Quill William Morrow and Company, Inc. 1991.

Rappley MD. Attention deficit-hyperactivity disorder. N Engl J Med. 2005;352:165–173.

Raz, N., Torres, I.J., Briggs, S.D., Spencer, W.D., Thornton, A.E., Loken, W.J., Gunning, F.M., McQuain, J.D., Driesen, N.R., Acker, J.D. 1995. Selective neuroanatomic abnormalities in Down's syndrome and their cognitive correlates: evidence from MRI morphometry. Neurology. 45, 356–366.

Reed HE, McGrew SG, Artibee K, Surdkya K, Goldman SE, Frank K, Wang L, Malow BA. Parent-Based Sleep Education Workshops in Autism. J Child Neurol. 2009;24(8):936-45.

Richdale AL, Prior MR. The sleep/wake rhythm in children with autism. Eur Child Adolesc Psychiatry. 1995;4(3):175-86.

Richdale AL. Sleep problems in autism: prevalence, cause, and intervention. Dev Med Child Neurol. 1999;41(1):60-6

Ring A, Stein D, Barak Y, Teicher A, Hadjez J, Elizur A, et al. Sleep disturbances in children with attention-deficit/hyperactivity disorder: a comparative study with healthy siblings. J Learn Disabil. 2000;31:572-8.

Rodopman-Arman A, Perdahli-Fiş N, Ekinci O, Berkem M. Sleep habits, parasomnias and associated behaviors in school children with attention deficit hyperactivity disorder (ADHD). Turk J Pediatr. 2011;53(4):397-403.

Rodrigue JR, Morgan SB, Geffken GR. 1991. A comparative evaluation of adaptive behavior in children and adolescents with autism, Down syndrome, and normal development. Journal of Autism and Developmental Disorders 1991;21:187–196. [PubMed: 1830878]

Roizen NJ, Patterson D. 2003. Down's syndrome. Lancet. 361:1281-1289

Romanos M, Gerlach M, Warnke A, Schmitt . Association of attention-deficit/hyperactivity disorder and atopic eczema modified by sleep disturbance in a large population-based sample. J Epidemiol Community Health. 2010; 64:269-273.

Rossignol DA, Frye RE. Melatonin in autism spectrum disorders: a systematic review and meta-analysis. Dev Med Child Neurol. 2011;53(9):783-92.

Rubenstein, J.L., Merzenich, M.M., 2003. Model of autism: increased ratio of excitation/inhibition in key neural systems. Genes Brain Behav. 2, 255–267.

Rueda N, Florez J, Martinez-Cue C. 2008. Effects of chronic administration of SGS-111 during adulthood and during the pre- and post-natal periods on the cognitive deficits of Ts65Dn mice, a model of Down syndrome. Behav, Brain Res. 188: 355–367.

Sahin U, Ozturk O, Ozturk M, Songur N, Bircan A, Akkaya A. Habitual snoring in primary school children: prevalence and association with sleep-related disorders and school performance. Med Princ Pract. 2009;18(6):458-65.

Sakamoto T, Cansev M, Wurtman RJ. 2007. Oral supplementation with docosahexaenoic acid and uridine-5´-monophosphate increases dendritic spine density in adult gerbil hippocampus. Brain Res. 1182:50-59.

Sakamoto T, Cnsev M, Wurtman, R.J. 2007. Oral supplementation with docosahexaenoic acid and uridine-5'-monophospate increases dendritic spine density in adult gerbil hippocampus. Brain Res. 50-59.

Salas C, Cambianica I, Rossi F. 2008. Molecular mechanisms of dendritic spine development and maintenance. Acta Neurobiol. Exp. 68:289-304.

Schalock, R., Snell, m., Spitalnik, D., Retraso Mental: Definición, clasificación y sistemas de apoyo (traducción de M. A. Verdugo y C. Jenaro), Madrid, Alianza Editorial, 1997

Schalock, R. y Verdugo, M.A., Calidad de vida. Manual para de la educación, salud y servicios sociales. Madrid, Alianza Editorial, 2003.

Scheweitzer JB, Cummins TK, Kant CA. Attention deficit/hyperactivity disorder. Med Clin North Am. 2001;85:755-77.

Schmidt, Michael A. (1997). "Smart Fats: How dietary fats and oils affect mental, physical and emotional intelligence". North Atlantic Books.

Schnoll R, Burshteyn D, Cea-Aravena J. Nutrition in the treatment of attention-deficit hyperactivity disorder: a neglected but important aspect. Appl Psychophysiol Biofeedback. 2003; 28:63–75.

Schwartz G, Amor LB, Grizenko N, Lageix P, Baron C, Boivin DB, et al. Actigraphic monitoring during sleep of children with ADHD on methylphenidate and placebo. J Am Acad Child Adolesc Psychiatry. 2004;43:1276-82.

Sciberras E, Efron D, Gerner B, Davey M, Mensah F, Oberklaid F, Hiscock H. Study protocol: the sleeping sound with attention-deficit/hyperactivity disorder project. BMC Pediatr. 2010:30;10:101.

Sciberras E, Fulton M, Efron D, Oberklaid F, Hiscock H. Managing sleep problems in school aged children with ADHD: A pilot randomised controlled trial. Sleep Med. 2011;12(9):932-5.

Secretaría de Comercio y Fomento Industrial y Secretaría de Salud de los Estados Unidos Mexicanos. NORMA Oficial Mexicana NOM-051-SCFI/SSA1-2010, Especificaciones

generales de etiquetado para alimentos y bebidas no alcohólicas preenvasados-Información comercial y sanitaria. 2010. México. Disponible en: http://dof.gob.mx/nota\_detalle\_popup.php?codigo=5137518

Secretaría de Salud de los Estados Unidos Mexicanos. Norma Oficial Mexicana NOM-086-SSA1-1994, Bienes Y Servicios. Alimentos Y Bebidas No Alcoholicas Con Modificaciones En Su Composicion. Especificaciones Nutrimentales. 1994. México. Disponible en: http://www.salud.gob.mx/unidades/cdi/nom/086ssa14.html

Secretaría de Salud. Gobierno Federal de los Estados Unidos Mexicanos. "NORMA Oficial Mexicana NOM-008-SSA2-1993, Control de la nutrición, crecimiento y desarrollo del niño y del adolescente. Criterios y procedimientos para la prestación del servicio." 1994. Disponible en: www.salud.gob.mx/unidades/cdi/nom/008ssa23.html

Secretaría de Salud. Gobierno Federal de los Estados Unidos Mexicanos. "NORMA Oficial Mexicana NOM-174-SSA1-1998, Para el manejo integral de la obesidad." Disponible en: http://www.salud.gob.mx/unidades/cdi/nom/174ssa18.html

Sekine, Kasunori; Watanabe-Sekine, Emiko; Toida, Tomohiro; Kahashima, Takuji; Kataoka, Tateshi; Hashimoto, Yoshiyuki. (1994) "Adjuvant Activity of the Cell Wall of Bifidobacterium infantis for in vivo Immune Responses in Mice". Immunopharmacol Immunotoxicol, Vol 16, 589-609.

Disponible en: http://informahealthcare.com/doi/abs/10.3109/08923979409019741

Sekine, Kazunori; Kahashima, Takuji & Hashimoto, Yoshiyuki. (1994). "Comparison of the TNF-α Levels Induced by Human-Derived Bifidobacterium longum and Rat-Derived Bifidobacterium animalis in Mouse Peritoneal Cells". Bifidobacteria Microflora. Vol 13, 79-89. Disponible en: https://www.jstage.jst.go.jp/article/bifidus1982/13/2/13\_2\_79/\_pdf

Sekine, Kazunori; Ohta, Jun; Onishi, Masatoshi; Tatsuki, Taro; Shimokawa, Yukiko; Toida, Tomohiro; Takuji, Kawashima & Yoshiyuki, Hashimoto (1995) "Analysis of Antitumor Properties of Effector Cells Stimulated With a Cell Wall Preparation (WPG) of Bifidobacterium Infantis". Biological and Pharmaceutical Bulletin, Vol 18, 148-153. Disponible en: https://www.jstage.jst.go.jp/article/bpb1993/18/1/18\_1\_148/\_pdf

Seltzer MM, Krauss MW, Shattuck PT, Orsmond G, Swe A, Lord C. 2003. The symptoms of autism spectrum disorders in adolescence and adulthood. Journal of Autism and Developmental Disorders 2003;33:565–581. [PubMed: 14714927]

Sergeant JA, Oosterlaan J, Van Der Meere J. Information processing in attention-deficit/hyperactivity disorder. En: Quay HC, Hogan AE, editors. Handbook of disruptive behavior disorders. New York: Plenum Press; 1999. p. 75-104.

Shaw William, Ph D., Autism Beyond the Basics, Kansas 2009.

Shaw William, PhD., Tratamientos Biológicos del Autismo y TDA, Kansas. 2006.

Shaw, William (2008). "Biological Treatments for Autism & PDD. Causes and Biomedical Therapies for Autism and PDD". 3<sup>a</sup> edición. U.S.A. Disponible en: http://www.greatplainslaboratory.com/home/eng/drshawbook.asp

Shaw, Willian. 2008. Biological Treatments for Autism and PDD. 3rd Revision. EEUU. http://www.biologicaltreatments.com/book/ch1.asp

Shen M, Hoogenraad CC. 2007. The postsynaptic architecture of excitatory synapses: a more quantitative view. Ann. Rev. Biochem. 76:823-847.

Sherman SL, Allen EG, Bean LH, Freeman SB. 2007. Epidemiology of Down syndrome. Mental Retar. Develop. Dis. Res. Rev. 13: 221-227.

Sheveli M, Schreiber R. Pemoline-associated hepatic failure: a critical analysis of the literature. Pedriatr Neurol. 1997;16:14-6.

Sigman M, Ruskin E. 1999. Continuity and change in the social competence of children with autism, Down syndrome, and developmental delays. Monographs of the Society for Research in Child Development 1999;64(1, Serial No. 256):v–114.

Silvestri R, Gagliano A, Arico I, Calesse, Cedro, Bruni O, Concluso R, Germano E, Gennovi G, Siracusano R, Vita G, Bramante P. Sleep dissorders in children with attention-deficit/hyperactivity disorder (ADHD) recorded overnight by video-polysomnography. Sleep Med. 2009;10(10):1132-8.

Sinn N, Bryan J, Wilson C. Cognitive effects of polyunsaturated fatty acids in children with attention deficit hyperactivity disorder symptoms: a randomized controlled trial. Prostaglandins Leukot Essent Fatty Acids. 2008;78:311–326.

Sinn N. Nutritional and dietary influences on attention deficit hyperactivity disorder. Nutr Rev. 2008;66:558–568.

Sivertsen B, Posserud MB, Gillberg C, Lundervold AJ, Hysing M. Sleep Problems in Children With Autism Spectrum Problems: A Longitudinal Population-Based Study. Autism. 2011;8.

Smalley SL. Genetic influences in childhood-onset psychiatric disorders: autism and attention deficit/hyperactivity disorder. Am J Hum Genet. 1997;60:1276-82.

Smith KM, Daly M, Fisher M, Yiannoutsos CT, Bauer L, Barkley R, et al. Association of the dopamine beta hydroxylase gene with attention deficit disorder: genetic analysis of the Milwaukee longitudinal study. Am J Med Genet. 2003;15:77-85.

Sonnenberg, Amnon & Müller, Astrid D. (1993). "Constipation and Cathartics as Risk Factors of Colorectal Cancer: A Meta-Analysis". División de Gastroenterología, de la Universidad de Wisconsin, Milwakee, EEUU. Pharmacology, International Journal of Experimental and Clinical Pharmacology. Volume 47, Supplement 1, 224-233.

Sonuga-Barke EJ. Psychological heterogeneity in AD/HD-a dual pathway model of behaviour and cognition. Behav Brain Res. 2002;130:29-36.

Souders MC; Mason TBA; Valladares O; Bucan M; Levy SE; Mandell DS; Weaver TE; Pinto-Martin D. Sleep behaviors and sleep quality in children with autism spectrum disorders. Sleep 2009;32(12):1566-1578.

Squire LR, Wixted JT, Clark RE. 2007. Recognition memory and the medial temporal lobe: a new perspective. Nat. Rev. Neurosci. 8(11): 872–883.

Starobrat-Hermelin B, Kozielec T. The effects of magnesium physiological supplementation on hyperactivity in children with attention deficit hyperactivity (ADHD). Positive response to magnesium oral loading test. Magnes Res. 1997;10:149–156.

Stein MA. Unrevealling sleep problems in treated and untreated children with ADHD. J Child Adolesc Psychopharmacol. 1999;9:157-68.

Stoll C, Alembik Y, Dott B, Roth MP, 1990. Epidemiology of Down syndrome in 118,265 consecutive births. Am. J. Med. Genet. 7 (Suppl.): 79–83.

Suetsugu M, Mehraein P. 1980. Spine distribution along the apical dendrites of the pyramidal neurons in Down's syndrome. A quantitative study. Acta Neuropathol. 50: 207-210.

Sung V, Hiscock H, Sciberras E, Efron D. Sleep problems in children with attention-deficit/hyperactivity disorder: prevalence and the effect on the child and family. Arch Pediatr Adolesc Med. 2008;162(4):336-42.

Suzuki, Ykio; Uchida, Kei. (1992). "Formation of β-Fructosyl Compounds of Pyridoxine in Growing Culture of Aspergillus niger". Instituto de Investigación de Biorecursos de la Universidad de Okayama, Japón. Bioscience, Biotechnology & Biochemistry Journal, Vol 57, Issue 6, 875-880. Disponible en: https://www.jstage.jst.go.jp/article/bbb1992/57/6/57\_6\_875/\_pdf

Swanson JM, Flodman P, Kennedy J, Spence MA, Moyzis R, Schuck S, et al. Dopamine genes and ADHD. Neurosci Biobehav Rev. 2000;24:21-5.

Tahiri, Maha; Tressol, JC; Arnaud, Josaine, Bornet, Francis; Bouteloup-Demange, Corinne; Feillet-Coudray, C. (2001) "Five week intake of short-chain fructooligosaccharides

increases intestinal absorption and status of magnesium in postmenopausal women". Journal of Bone Mineral Research. Vol 16, Issue 11, 2152-2160.

Tahiri, Maha; Tressol, Jean C; Arnaud, Jaosaine; Bornet, Francis RJ; Bouteloup-Demange, Corinne; Feillet-Coudray, Christine; Brandolini, Marion; Ducros, Véronique; Pépin, Denise; Brouns, Fred; Roussel, Anne Marie; Rayssiguier, Yves & Coudray, Charles. (2003). "Effect of short-chain fructooligosaccharides on Intestinal Calcium Absorption and Calcium Status in Postmenopausal Women: A Stable-Isotope Study". The American Journal of Clinical Nutrition. Vol 77, No 2, 449-457. Disponible en: http://www.ajcn.org/content/77/2/449.full.pdf+html

Takashima S, Becker L, Armstrong DL, Chan F. 1981. Abnormal neuronal development in the visual cortex of the human fetus and infant with Down's syndrome. A quantitative and qualitative golgi study. Brain Res. 225: 1-21.

Tannock R. Attention deficit hyperactivity disorder: advances in cognitive, neurobiological and genetic research. J Child Psychol Psychiatry. 1998;39:65-99.

Tasker A, Dettmar PW, Panetti M, Kourman JA, Birchall JP, Pearson JP. Reflux of gastric juice and glue ear in children. Lancet. 2004;359:493.

Ting H, Wong RH, Yang HJ, Lee SP, Lee SD, Wang L. Sleep-disordered breathing, behavior, and academic performance in Taiwan schoolchildren. Sleep Breath. 2011;15(1):91-8.

Tininenko JR ,Fisher PA, Bruce J, Pears KC. Associations Between Sleep and Inattentive/Hyperactive Problem Behavior Among Foster and Community Children. J Dev Behav Pediatr. J Dev Behav Pediatr. 2010;31(8):668-74.

Tirosh E, Sadeh A, Munvez R, Lavie P. Effects of methylphenidate on sleep in children with attention-deficit hyperactivity disorder. Am J Dis Child. 1993;147:1313-5. 76.

Todd RD, Botteron KN. Is attention-deficit/hyperactivity disorder an energy deficiency syndrome? Biol Psychiatry. 2001;50:151-8.

Tomás Vila M, Miralles Torres A, Beseler Soto B. Versión española del Pediatric Sleep Questionnaire. Un instrumento útil en la investigación de los trastornos del sueño en la infancia. Análisis de su fiabilidad. An Pediatr (Barc). 2007;66:121-8.

Touchette E, Côté SM, Petit D, Liu X, Boivin M, Falissard B, Tremblay RE, Montplaisir JY. Short Nighttime Sleep-Duration and Hyperactivity Trajectories in Early Childhood. Pediatrics. 2009;124(5):985-993

Turkel H. Medical amelioration of Down's syndrome incorporating the orthomolecular approach. Journal of Orthomolecular Psychiatry, 4:102-115, 1975.

U.S. Department of Health and Human Services. Healthy People 2010: Understanding and Improving Health. 2nd. Washington, DC: U.S. Government Printing Office; Nov. 2000

Vaillend C, Poirier R, Laroche S. 2008. Genes, plasticity and mental retardation. Behav. Brain Res. 192(1):88 105.

Vallabhajosula, S; Goldsmith, SJ; Lipszyc, H & Chahinian, AP. (1983). "67Ga-transferrin and 67Ga-lactoferrin binding to tumour cells: specific versus nonspecific glycoprotein-cell interaction". European Journal of Nuclear Mededicine. Volume 8, 354-357.

Varoqueaux, F., Aramuni, G., Rawson, R.L., Mohrmann, R., Missler, M., Gottmann, K., Zhang, W., Südhof, T.C., Brose, N., 2006. Neuroligins determine synapse maturation and function. Neuron 51, 741–754.

Vila MT. Efecto del metilfenidato sobre el sueño. Resultados de un estudio multicéntrico en una población infantil afecta de trastorno por déficit de atención e hiperactividad. An Pediatr (Barc). 2010.doi:10.1016/j.anpedi.2010.05.013

Vila MT. Torres AM. Soto BB. Gomar MR. Sala MJ. Al Sierra U. Relación entre el trastorno por déficit de atención e hiperactividad y los trastornos del sueño. Resultados de un estudio epidemiológico en la población escolar de la ciudad de Gandía. An Pediatr (Barc), 2008;69(3):251-7.

Vriend JL, Corkum PV, Moon EC, Smith IM. Behavioral Interventions for Sleep Problems in Children With Autism Spectrum Disorders: Current Findings and Future Directions. J. Pediatr Psychol. 2011; 36: 1017 1029.

Wagner ML, Walters AS, Fisher BC. Symptoms of attention-deficit/hyperactivity disorder in adults with restless legs syndrome. Sleep. 2004;27:1499-504.

Walters AS, Mandelbaum DE, Lewin DS, Kugler S, England SJ, Miller M. Dopaminergic therapy in children with restless legs/periodic limb movements in sleep and ADHD. Pediatr Neurol. 2000;22:182-6.

Wang, YZ; Xu CL; An, ZH; Liu, LX & Feng J. (2006). "Effect of Dietary Bovine Lactoferrin on Performance and Antioxidant Status of Piglets". Laboratorio de nutrición animal molecular de la Universidad de Zhejiang China.

Wang, Ze-Jian; Liang, Cui-Ling; Li, Guang-Mei; Yu, Cai-Yi & Yin, Ming. (2006). "Neuroportective effects of Arachidonic Acid Against Oxidative Stress on Rat Hippocampal Slices". Chemico-Biological Interactions. Volume 163, Issue 3, 207-217

Ward, Loren. (2006). "Lactoferrin Immune Enhancement and Prebiotic Activity". Glanbia Nutritionals.

Ward, Loren. (2006). "The Physiological Significance of Milk Minerals". Glanbia Foods inc.

Ward, Loren. (2007) "TruCAL Milk Calcium Significantly Increases Bone Strength and Improves Bone Biomarkers In Vivo" Glanbia Nutritionals Inc.

Wei JL, Bond J, Mayo MS, Smith HJ, Reese M, Weatherly RA. Improved Behavior and Sleep After Adenotonsillectomy in Children With Sleep-Disordered Breathing: Long-term Follow-up. Arch Otolaryngol Head Neck Surg. 2009;135:642-646.

Weiskop S, Richdale A, Matthews J. Behavioural treatment to reduce sleep problems in children with autism or fragile X syndrome. Dev Med Child Neurol. 2005;47(2):94-104

West CD, Kemper TL. 1976. The effect of a low protein diet on the anatomical development of the rat brain. Brain Res. 107: 221-237.

White D, Kaplitz SE. Treatment of Down's syndrome with a vitamin-mineral preparation. International Copenhagen Congress of the Scientific Studies of Mental Retardation 1:224-228, 1964.

Willoughby MT. Developmental course of ADHD symptomatology during the transition from childhood to adolescence: a review with recommendations. J Child Psychol Psychiatry. 2003;44:88-106.

Wirojanan J, Jacquemont S, Diaz R, Bacalman S, Anders TF, Hagerman RJ, Goodlin-Jones BL. The Efficacy of Melatonin for Sleep Problems in Children with Autism, Fragile X Syndrome, or Autism and Fragile X Syndrome. J Clin Sleep Med.2009;5(2):145-150.

Wisniewski KE, Schmidt-Sidor B. 1989. Postnatal delay of myelin formation in brains from Down syndrome infants and children. Clin. Neuropathol. 8: 55-62.

Wisniewski KE. 1990. Down syndrome children often have brain with maturation delay, retardation of growth, and cortical dysgenesis. Am. J. Genet. Suppl. 7: 274-281.

World Health Organization. The Tenth Revision of the International Classification of Diseases and related health problems (ICD-10). Geneve: WHO; 1992.

World Health Organization. WHO Reference 2001. "Growth reference data for 5 – 19 years old". Disponible en: http://www.who.int/growthref/en/

Wright B, Sims D, Smart S, Alwazeer A, Alderson-Day B, Allgar V, Whitton C, Tomlinson H, Bennett S, Jardine J, McCaffrey N, Leyland C, Jakeman C, Miles J. Melatonin Versus Placebo in Children with Autism Spectrum Conditions and Severe Sleep Problems Not Amenable to Behaviour Management Strategies: A Randomised Controlled Crossover Trial. J Autism Dev Disord. 2011;41(2):175-84.

Yasui Hisako; Nagoaka, N.; Mike, A.; Hayakawa, K.& Ohwaki, M. (1992) "Detection of Bifidobacterium Strains That Induce Large Quantities of IgA". Yakult Central Institute for Microbiological Research. Microbioal Ecology in Health and Diseases. Vol 5, 155-162. Japón. Disponible en: http://www.microbecolhealthdis.net/index.php/mehd/article/view/7838

Yasui, Hisako; Ohwaki, M. (1991). "Enhancement of Immune Response in Peyer's Parch Cells Cultured With Bifidobacterium Breve". Yakult Central Institute for Microbiological Research. Journal of Dairy Science Vol 74, Issue 1, 187-195. Japon. Disponible en: http://download.journals.elsevierhealth.com/pdfs/journals/0022-0302/PIIS0022030291782726.pdf

Yilmaz K, Kilincaslan A, Aydin N, Kor D. Prevalence and correlates of restless legs syndrome in adolescents. Dev Med Child Neurol. 2011; 53(1): 40-7.

Zhou Q, Homma KJ, Poo MM. 2004. Shrinkage of dendritic spine associated with long-term depression of hippocampal synapses. Neuron. 44: 749-757.

Ziv NE, Smith SJ. 1996. Evidence for a role of dendritic filopodia in synaptogenesis and spine formation. Neuron. 17(1):91-102.

# **APPENDIX "A": INFORMED CONSENT**

### ETHICAL CONSIDERATIONS AND/OR INFORMED CONSENT FORM

The principles of this informed consent process are grounded in the ethical foundations of the Declaration of Helsinki, the International Conference on Harmonization (ICH), Good Clinical Practice (GCP) guidelines, and all applicable regulatory requirements.

For this study, written informed consent will be obtained prior to the initiation of any procedure or evaluation by the investigator or an authorized delegate, as documented on the Delegation of Responsibilities Sheet.

Legal guardians of participants will be provided with both oral and written information regarding the nature and objectives of the study, as well as the procedures involved, before consent is obtained.

### INFORMED CONSENT TO PARTICIPATE IN A RESEARCH STUDY

**Protocol Title:** Neuro-Nutrition as Support for Physiological Performance and Cognitive Skills in Individuals with Trisomy 21, Autism Spectrum Disorders, and Attention Deficit Disorder.

| CONACYT Pro | ject Number: _ |
|-------------|----------------|
|-------------|----------------|

#### **Research Team:**

- Sleep Physiology Area Lead: Dr. Elizabeth Ibarra Coronado
- Biomedical Area Lead: I.B. Cecilia Fernández Aguirre
- Ethnographic Area Lead: Lic. Arturo Ramírez Ramos

### The study will be conducted at the following locations:

- DOMUS Instituto de Autismo
- Integración Down I.A.P.
- Facultad de Psicología Universidad Nacional Autónoma de México (UNAM)
- Instituto Mexicano de Medicina Integral de Sueño
- Participants' homes

| Name of Participant: |
|----------------------|
| • |

You and your child are invited to participate in this research study. Before making a decision, you should carefully read and understand each section of this document. This process is known as informed consent. Please feel free to ask any questions at any time to clarify any doubts you may have.

If you agree for your child to take part in the study, you will be asked to sign this consent form.

## JUSTIFICATION OF THE STUDY

Improvements in cognitive skills and overall quality of life have been documented in individuals with Down Syndrome (DS), Autism Spectrum Disorders (ASD), and Attention Deficit Disorders (ADD/ADHD) when dietary modifications eliminate gluten and casein and

incorporate nutritional supplements. The objective of this project is to extend these benefits to a broader population with the same conditions.

A maximum of 90 participants will be enrolled, each assigned to one of three groups (two dietary intervention groups and one control group) and monitored over the course of one year.

Progress will be evaluated through a combination of traditional laboratory tests (hematology, blood chemistry, cortisol, homocysteine, C-reactive protein, stool analyses), cognitive and behavioral assessments, polysomnography, event-related potentials (P300), anthropometric measurements, and ethnographic interviews. Additionally, specialized analyses will be performed in the United States, including Organic Acid Profile, IgG Food Allergy and Sensitivity Tests, and Gluten/Casein Peptide Assays.

#### **OBJECTIVE OF THE STUDY**

The purpose of this study is to investigate behavioral and cognitive changes in individuals with Autism Spectrum Disorders (ASD), Attention Deficit Disorder (ADD/ADHD), or Down Syndrome (DS) through dietary modification. The intervention specifically involves eliminating harmful dietary components while incorporating nutrients that are typically under-metabolized due to the underlying characteristics of these conditions.

#### **BENEFITS OF THE STUDY**

The study aims to expand scientific knowledge on the role of nutrition in cognitive functioning among individuals with these conditions, with the goal of supporting therapeutic management and contributing to the improvement of quality of life.

### **STUDY PROCEDURES**

If you consent for your child to participate, the following procedures will be performed:

- Blood, urine, and stool tests.
- Medical examinations by specialists.
- Cognitive and behavioral assessments.
- Ethnographic interviews and questionnaires.
- Polysomnographic sleep studies to evaluate sleep physiology.

These procedures are non-invasive and will not cause pain.

### RISKS ASSOCIATED WITH THE STUDY

No significant risks are expected from the procedures mentioned.

#### **CLARIFICATIONS**

- Participation is voluntary.
- All dietary guidelines, supplement intake, and dosage instructions must be followed precisely.
- Parents are required to attend support sessions throughout the research period.
- Declining participation will not result in any negative consequences.
- You may withdraw your child at any time without penalty by informing the research team.
- There will be no cost to you for the tests or procedures required for this study.
- No financial compensation will be provided for participation.
- Confidentiality of personal and medical information will be strictly maintained.
- If participation requirements (dietary compliance, supplement intake) are not met, the research team may ask you to withdraw without prejudice.
- Periodic progress reports will be provided to participating families during the study.

If you agree to participate, you formally commit to complying with the nutritional instructions provided, as these are essential for the accuracy and validity of the study results.

| INFORMED CONSENT FORM | | | |
|---|---|---|---|
| l, | , have | e read and understood the informat | on |
| above, and my questions have b | been answered | d satisfactorily. I understand that st | udy data |
| may be used for scientific purpo | oses. I consen | t to participate in this research stud | у. |
| Parent/Guardian Signature: _ | | Date: | |
| Witness: | Date: | | |

| Witness: | Date: |
|---|---|
| Investigator's Statement: I have explained to Mr./Ms the nature and purpose of the research, the risks and benefits of participation, and answered questions to the best of my ability. I certify that I am familiar with applicable ethical standards for research involving human participants. | |
| Investigator's Signature: | Date: |
| CONSENT WITHDRAWAL FORM | |
| | hase II as Support for Physiological Performance and<br>Trisomy 21, Autism Spectrum Disorders, and Attention |
| <b>Study Sites</b> The study will be conducted at the | e following locations: |
| DOMUS Instituto de Autisn | mo |
| • Facultad de Psicología – U | niversidad Nacional Autónoma de México (UNAM) |
| Instituto Mexicano de Med | icina Integral de Sueño |
| <ul> <li>Participants' homes</li> </ul> | |
| Participant's Name: | |
| I hereby inform you of my voluntar<br>the following reasons: | ry decision to withdraw from this research protocol for |
| commit to returning any unused for | study information or documents will be provided, and I ormulation to the principal investigator. |
| Parent/Guardian Signature: | Date: |
| Witness: | Date: |
| Witness: | Date: |